CLINICAL TRIAL: NCT02304367
Title: A Phase 2 Open-Label Trial to Assess the Efficacy and Safety of KRN23, an Antibody to FGF23, in Subjects With Tumor-Induced Osteomalacia (TIO) or Epidermal Nevus Syndrome (ENS)-Associated Osteomalacia
Brief Title: Study of Burosumab (KRN23) in Adults With Tumor-Induced Osteomalacia (TIO) or Epidermal Nevus Syndrome (ENS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin, Inc. (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UX023T-CL201
Expanded Access: NCT03775187 (Available)
Record Dates: First submitted 2014-11-24; First posted 2014-12-01 (Estimated); Results first posted 2020-07-30 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Tumor Induced Osteomalacia (TIO); Epidermal Nevus Syndrome (ENS)
Keywords: TIO; ENS; FGF23; KRN23
MeSH Terms: conditions — Oncogenic osteomalacia; Nevus, Sebaceous of Jadassohn | interventions — burosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Burosumab (Experimental): Participants received burosumab at a starting dose of 0.3 mg/kg administered subcutaneously (SC) every 4 weeks (Q4W). Doses may have been titrated up to a maximum of 2.0 mg/kg every 2 weeks (Q2W) in order to achieve fasting peak serum phosphorus levels within the target range of 2.5 to 4.0 mg/dL.
  Interventions: Biological: Burosumab

INTERVENTIONS:
Biological: Burosumab — Solution for subcutaneous injection
  Other Names: KRN23; Crysvita®; UX023

SUMMARY:
The primary objectives of this study are to evaluate the effect of burosumab treatment on:

* Increasing serum phosphorus levels in adults with TIO or ENS-associated osteomalacia
* Improvement in TIO/ENS-associated osteomalacia as determined by osteoid thickness (O.Th), osteoid surface/bone surface (OS/BS), osteoid volume/bone volume (OV/BV) and mineralization lag time (MLt).

ELIGIBILITY:
Inclusion Criteria:

1. Have a clinical diagnosis of TIO/ENS-associated osteomalacia based on evidence of excessive fibroblast growth factor 23 (FGF23) that was not amenable to cure by surgical excision of the underlying tumor/lesion (documented by Investigator).
2. Be ≥ 18 years of age
3. Have a fasting serum phosphorus level < 2.5 mg/dL
4. Have an FGF23 level ≥ 100 pg/mL by Kainos assay
5. Have a ratio of renal tubular maximum reabsorption rate of phosphate to glomerular filtration rate (TmP/GFR) < 2.5 mg/dL
6. Have an estimated glomerular filtration rate (eGFR) ≥ 60 mL/min (using Cockcroft-Gault formula). Subjects with eGFR ≥ 30 but < 60 mL/min will be considered eligible as long as in the opinion of the investigator the decline in renal function is not related to nephrocalcinosis.
7. Have a corrected serum calcium level < 10.8 mg/dL
8. Females of child-bearing potential must have a negative urine pregnancy test at Screening and Baseline and be willing to have additional pregnancy tests during the study. Females considered not to be of childbearing potential include those who have not experienced menarche, are post-menopausal (defined as having no menses for at least 12 months without an alternative medical cause) or are permanently sterile due to total hysterectomy, bilateral salpingectomy, or bilateral oophorectomy.
9. Be willing to use 2 forms of effective methods of contraception while participating in the study (sexually active subjects) and for 12 weeks after last dose of study drug.
10. Be willing to provide access to prior medical records to determine eligibility including imaging, biochemical, and diagnostic, medical, and surgical history data
11. Provide written informed consent after the nature of the study has been explained, and prior to any research-related procedures
12. Be willing and able to complete all aspects of the study, adhere to the study visit schedule and comply with the assessments (in the opinion of the investigator)

Exclusion Criteria:

1. Have a prior diagnosis of human immunodeficiency virus (HIV), hepatitis B and/or hepatitis C
2. Have a history of recurrent infection, a predisposition to infection, or a known immunodeficiency
3. Are pregnant or breastfeeding at Screening or are planning to become pregnant (self or partner) at any time during the study
4. Have participated in an investigational drug or device trial within 30 days prior to Screening or are currently enrolled in another study of an investigational product or device
5. Have used a therapeutic monoclonal antibody (mAb), including KRN23, within 90 days prior to Screening or have a history of allergic or anaphylactic reactions to any mAb
6. Have or a have a history of any hypersensitivity to KRN23 excipients that, in the judgment of the investigator, places the subject at increased risk for adverse effects
7. Have used a pharmacologic vitamin D metabolite or its analog (e.g., calcitriol, doxercalciferol, and paricalcitol), phosphate, or aluminum hydroxide antacids (e.g., Maalox® and Mylanta®) within 2 weeks prior to Screening or during the study
8. Have used medication to suppress parathyroid hormone (PTH) (e.g., Sensipar®, cinacalcet, calcimimetics) within 2 months prior to Screening
9. Have a history of malignancy within 5 years of study entry with the exception of phosphaturic mesenchymal tumors (PMTs) of the mixed connective tissue type or non-melanoma skin cancers such as basal cell skin cancer
10. Have donated blood or blood products within 60 days prior to Screening
11. Have a history of allergic reaction to or have shown adverse reactions to a tetracycline (e.g., tetracycline hydrochloride [HCl] and demeclocycline), benzodiazepines, fentanyl or lidocaine
12. Have any condition, which in the opinion of the investigator and sponsor, could present a concern for either subject safety or difficulty with data interpretation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-03-24 (Actual); Primary Completion 2017-07-27 (Actual); Study Completion 2021-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (7):
- United States (7):
  - Colorado Center for Bone Research at Panorama Orthopedics and Spine Center, Golden, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Indiana University Hospital, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Duke University, Durham, North Carolina
  - Houston Methodist Research Institute, Houston, Texas

REFERENCES:
- [Derived] Khadora M, Mughal MZ. Burosumab treatment in a child with cutaneous skeletal hypophosphatemia syndrome: A case report. Bone Rep. 2021 Oct 1;15:101138. doi: 10.1016/j.bonr.2021.101138. eCollection 2021 Dec. PMID 34660853

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 8 centers in the United States, and enrolled adults with tumor-induced osteomalacia (TIO), epidermal nevus syndrome (ENS)-associated osteomalacia, or x-linked hypophosphatemia (XLH).
Period: Overall Study
Arm/Group | Burosumab
Started | 17 (14 participants with TIO; 1 participant with ENS; 2 participants with XLH)
Completed 48 Weeks of Study Drug | 16
Completed 144 Weeks of Study Drug | 12
Completed | 9
Not Completed | 8
Not completed — Lack of Response to Bruosumab | 1
Not completed — Sponsor Decision | 3
Not completed — Death | 2
Not completed — Physician Decision | 1
Not completed — Unable to Return Due to Corona Virus Pandemic | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Arm/Group | Burosumab
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (13.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Black or African American | 2
  Native Hawaiian or Other Pacific Islander | 0
  White | 15
  Other | 0
Diagnosis [Count of Participants; unit: Participants] — Two participants who were enrolled in the study with a clinical diagnosis of TIO were later found to have X-linked hypophosphatemia (XLH) based on genetic testing.
  Participants
    Tumor-Induced osteomalacia (TIO) | 14
    Epidermal nevus syndrome-associated osteomalacia | 1
    X-linked hypophosphatemia (XLH) | 2
Serum Total Fibroblast Growth Factor 23 (FGF23) [Mean (Standard Deviation); unit: pg/mL] — Population: Tumor-induced osteomalacia (TIO) analysis set includes the 14 participants with TIO who received at least 1 dose of study drug.
  pg/mL
    number analyzed (Participants) | 14
    (all) | 770.06 (797.654)
Serum Phosphorus [Mean (Standard Deviation); unit: mg/dL] — Population: TIO analysis set
  mg/dL
    number analyzed (Participants) | 14
    (all) | 1.60 (0.474)
Osteoid Volume/Bone Volume (OB/BV) [Mean (Standard Deviation); unit: percentage of bone volume] — The percentage of a given volume of bone tissue that consists of unmineralized bone (osteoid). Population: TIO biopsy analysis set includes 11 participants with TIO who received at least 1 dose of study drug and who had paired bone biopsies at Baseline and Week 48.
  percentage of bone volume
    number analyzed (Participants) | 11
    (all) | 17.61 (19.485)
Osteoid Surface/Bone Surface (OS/BS) [Mean (Standard Deviation); unit: percentage of bone surface] — The percentage of bone surface covered in osteoid. Population: TIO biopsy analysis set
  percentage of bone surface
    number analyzed (Participants) | 11
    (all) | 56.82 (31.003)
Osteoid Thickness (O.Th) [Mean (Standard Deviation); unit: μm] — Mean thickness, given in micrometers, for osteoid seams Population: TIO biopsy analysis set
  μm
    number analyzed (Participants) | 11
    (all) | 16.45 (12.044)
Mineralization Lag Time (Mlt) [Mean (Standard Deviation); unit: days] — Mineralization lag time is the average time interval between osteoid formation and its subsequent mineralization, calculated by dividing the osteoid width by the mineralizing apposition rate (MAR; the average rate at which new bone mineral is being added on any actively forming surface).
  If Mlt could not be calculated directly due to low tetracycline uptake, Mlt was imputed according to the following:
  Mlt = O.Th/(MAR*MS/OS), where O.Th = osteoid thickness, MAR is imputed as 0.3 μm/day, MS/OS=Mineralizing Surface/Osteoid Surface, each measured at the same visit. Population: TIO biopsy analysis set for whom Mlt could be calculated or imputed
  days
    number analyzed (Participants) | 10
    (all) | 1597.73 (1326.832)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Mean Serum Phosphorus Levels Above 2.5 mg/dL at the Mid-Point of the Dose Intervals Between Baseline and Week 24
Description: The percentage of participants achieving mean serum phosphorus levels above the lower limit of normal (LLN; 2.5 mg/dL [0.81 mmol/L]) at the mid-point of the dose interval (2 weeks after dosing), as averaged across dose cycles between Baseline and Week 24 (i.e. the average of serum phosphorus levels at Weeks 2, 6, 10, 14 and 22).
Time Frame: Mid-point of each dose interval from Baseline to Week 24 (Weeks 2, 6, 10, 14 and 22 [there was no study visit at Week 18])
Population: TIO analysis set: includes participants with TIO who received at least 1 dose of burosumab during the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Burosumab
Number analyzed (Participants) | 14
percentage of participants | 50.0 [26.80 to 73.20]

2. Primary Outcome: Change From Baseline to Week 48 in Osteoid Thickness
Description: Histomorphometry of trans-iliac crest bone biopsies was assessed by a blinded, central reader.
  Osteoid thickness is the mean thickness of osteoid seams.
Time Frame: Baseline, Week 48
Population: TIO bone biopsy analysis set
Measure: Mean (95% Confidence Interval); unit: µm
Arm/Group | Burosumab
Number analyzed (Participants) | 11
µm | -5.12 [-10.04 to -0.20]
Statistical Analysis 1: Comparison: Burosumab; The null hypothesis that the mean change from Baseline to Week 48 in osteoid thickness is zero was tested using a t-test; Test type: Other; p = 0.0428, t-test

3. Primary Outcome: Change From Baseline to Week 48 in Osteoid Surface/Bone Surface (OS/BS)
Description: Histomorphometry of trans-iliac crest bone biopsies was assessed by a blinded, central reader.
  Osteoid surface/bone surface is expressed as the percentage of bone surface covered in osteoid.
Time Frame: Baseline, Week 48
Population: TIO biopsy analysis set
Measure: Mean (95% Confidence Interval); unit: percentage of bone surface
Arm/Group | Burosumab
Number analyzed (Participants) | 11
percentage of bone surface | -0.18 [-13.86 to 13.50]
Statistical Analysis 1: Comparison: Burosumab; The null hypothesis that the mean change from Baseline to Week 48 in OS/BS is zero was tested using a t-test; Test type: Other; p = 0.9770, t-test

4. Primary Outcome: Change From Baseline to Week 48 in Osteoid Volume/Bone Volume (OV/BV)
Description: Histomorphometry of trans-iliac crest bone biopsies was assessed by a blinded, central reader. Osteoid volume/bone volume is expressed as the percentage of a given volume of bone tissue that consists of unmineralized bone (osteoid).
Time Frame: Baseline, Week 48
Population: TIO bone biopsy analysis set
Measure: Mean (95% Confidence Interval); unit: percentage of bone volume
Arm/Group | Burosumab
Number analyzed (Participants) | 11
percentage of bone volume | -5.47 [-11.87 to 0.93]
Statistical Analysis 1: Comparison: Burosumab; The null hypothesis that the mean change from Baseline to Week 48 in OV/BV is zero was tested using a t-test; Test type: Other; p = 0.0858, t-test

5. Primary Outcome: Change From Baseline to Week 48 in Mineralization Lag Time (MLt)
Description: Mineralization lag time is a dynamic modeling parameter representing the mean time interval between the formation of osteoid and its subsequent mineralization which can be measured using histomorphometry with double tetracycline labeling.
  Mlt was calculated by dividing the osteoid width by the mineralizing apposition rate (MAR; the average rate at which new bone mineral is being added on any actively forming surface).
  If Mlt could not be calculated directly due to low tetracycline uptake, Mlt was imputed according to the following:
  Mlt = O.Th/(MAR*MS/OS), where O.Th = osteoid thickness, MAR is imputed as 0.3 μm/day, MS/OS=mineralizing surface/osteoid surface, each measured at the same visit.
Time Frame: Baseline, Week 48
Population: TIO biopsy analysis set for whom Mlt could be calculated or imputed
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Burosumab
Number analyzed (Participants) | 10
days | -565.20 [-2037.42 to 907.02]
Statistical Analysis 1: Comparison: Burosumab; The null hypothesis that the mean change from Baseline to Week 48 in Mlt is zero was tested using a t-test; Test type: Other; p = 0.4077, t-test

6. Secondary Outcome: Percentage of Participants Achieving Mean Serum Phosphorus Levels Above 2.5 mg/dL at the End of the Dose Intervals Between Baseline and Week 24
Description: The percentage of participants achieving mean serum phosphorus levels above the lower limit of normal (2.5 mg/dL [0.81 mmol/L]) at the end of the dose interval (4 weeks post-dose, prior to the next dose), as averaged across dose cycles between Baseline and Week 24 (i.e. the average of serum phosphorus levels at Weeks 4, 8, 12, 16, 20, and 24).
Time Frame: End of each dose interval from Baseline to Week 24 (Weeks 4, 8, 12, 16, 20, and 24)
Population: TIO analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Burosumab
Number analyzed (Participants) | 14
percentage of participants | 21.4 [7.57 to 47.59]

7. Secondary Outcome: Mean Change From Baseline in Serum Phosphorus Levels at the Mid-Point of the Dose Interval, as Averaged Across Dose Cycles Between Baseline and Week 24
Description: Mean change from Baseline to the mid-point of the dose interval (2 weeks after dosing) averaged across dose cycles between Baseline and Week 24 (i.e. the average of serum phosphorus levels at Weeks 2, 6, 10, 14 and 22).
Time Frame: Baseline and the mid-point of each dose interval from Baseline to Week 24 (Weeks 2, 6, 10, 14 and 22)
Population: TIO analysis set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Burosumab
Number analyzed (Participants) | 14
mg/dL | 1.039 (0.5622)

8. Secondary Outcome: Percent Change From Baseline in Serum Phosphorus Levels at the Mid-Point of the Dose Interval, as Averaged Across Dose Cycles Between Baseline and Week 24
Description: Mean percent change from Baseline to the mid-point of the dose interval (2 weeks after dosing) averaged across dose cycles between Baseline and Week 24 (i.e. the average of serum phosphorus levels at Weeks 2, 6, 10, 14 and 22).
Time Frame: Baseline and the mid-point of each dose interval from Baseline to Week 24 (Weeks 2, 6, 10, 14 and 22)
Population: TIO analysis set
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Burosumab
Number analyzed (Participants) | 14
percent change | 69.77 (43.743)

9. Secondary Outcome: Mean Change From Baseline in Serum Phosphorus Levels at the End of the Dosing Cycle, as Averaged Across Dose Cycles Between Baseline and Week 24
Description: Mean change from Baseline at the end of the dose interval (4 weeks post-dose, prior to the next dose) averaged across dose cycles between Baseline and Week 24 (i.e. the average of serum phosphorus levels at Weeks 4, 8, 12, 16, 20, and 24).
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, and 24
Population: TIO analysis set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Burosumab
Number analyzed (Participants) | 14
mg/dL | 0.550 (0.4260)

10. Secondary Outcome: Percent Mean Change From Baseline in Serum Phosphorus Levels at the End of the Dosing Cycle, as Averaged Across Dose Cycles Between Baseline and Week 24
Description: Mean percent change from Baseline at the end of the dose interval (4 weeks post-dose, prior to the next dose) averaged across dose cycles between Baseline and Week 24 (i.e. the average of serum phosphorus levels at Weeks 4, 8, 12, 16, 20, and 24).
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, and 24
Population: TIO analysis set
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Burosumab
Number analyzed (Participants) | 14
percent change | 38.56 (33.027)

11. Secondary Outcome: Time-Adjusted Area Under the Curve (AUC) of Serum Phosphorus Levels Between Baseline and Week 24
Description: Serum phosphorus level versus time AUC was calculated using the trapezoidal rule. Time-adjusted AUC was calculated by dividing the AUC by duration of time included in AUC calculation.
Time Frame: Pre-dose on Day 1 and at Weeks 1, 2, 4, 6, 8, 10, 12, 14, 16, 20, 21, 22, and 24
Population: TIO analysis set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Burosumab
Number analyzed (Participants) | 14
mg/dL | 2.36 (0.632)

12. Secondary Outcome: Change From Baseline Over Time in Serum 1,25-dihydroxyvitamin D (1,25(OH)2D) Concentration
Description: Least squares (LS) means and standard errors (SE) were estimated from a generalized estimation equation (GEE) model which includes the change from Baseline as the dependent variable, time as the categorical variable and adjusted for Baseline 1,25(OH)2D, with compound symmetry covariance structure.
Time Frame: Baseline and Weeks 24, 48, 96, 144, 168, 192, 216, and 240
Population: TIO analysis set participants with available data at Baseline and each time point.
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Burosumab
Number analyzed (Participants) | 11
pg/mL
  Week 24 | 9.90 (4.10)
  Week 48: number analyzed (Participants) | 10
  Week 48 | 10.49 (4.82)
  Week 96: number analyzed (Participants) | 9
  Week 96 | 4.28 (3.80)
  Week 144: number analyzed (Participants) | 9
  Week 144 | 3.15 (3.34)
  Week 168: number analyzed (Participants) | 8
  Week 168 | 4.91 (3.94)
  Week 192: number analyzed (Participants) | 8
  Week 192 | 0.67 (4.19)
  Week 216: number analyzed (Participants) | 5
  Week 216 | 9.78 (3.04)
  Week 240: number analyzed (Participants) | 5
  Week 240 | 6.56 (3.19)
Statistical Analysis 1: Comparison: Burosumab; Week 24; Test type: Other; p = 0.016, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline 1,25(OH)2D
Statistical Analysis 2: Comparison: Burosumab; Week 48; Test type: Other; p = 0.030, GEE model; [statistical method as in outcome 12, analysis 1]
Statistical Analysis 3: Comparison: Burosumab; Week 96; Test type: Other; p = 0.259, GEE model; [statistical method as in outcome 12, analysis 1]
Statistical Analysis 4: Comparison: Burosumab; Week 144; Test type: Other; p = 0.346, GEE model; [statistical method as in outcome 12, analysis 1]
Statistical Analysis 5: Comparison: Burosumab; Week 168; Test type: Other; p = 0.213, GEE model; [statistical method as in outcome 12, analysis 1]
Statistical Analysis 6: Comparison: Burosumab; Week 192; Test type: Other; p = 0.873, GEE model; [statistical method as in outcome 12, analysis 1]
Statistical Analysis 7: Comparison: Burosumab; Week 216; Test type: Other; p = 0.001, GEE model; [statistical method as in outcome 12, analysis 1]
Statistical Analysis 8: Comparison: Burosumab; Week 240; Test type: Other; p = 0.040, GEE model; [statistical method as in outcome 12, analysis 1]

13. Secondary Outcome: Change From Baseline Over Time in Total Serum Fibroblast Growth Factor 23 (FGF23) Concentration
Description: Total FGF23 included free FGF23 and FGF23 bound to burosumab. Least squares means and standard errors were estimated from a generalized estimation equation (GEE) model which includes the change from Baseline as the dependent variable, time as the categorical variable and adjusted for Baseline total FGF23, with compound symmetry covariance structure.
Time Frame: Baseline and Weeks 24, 48, 96, 144, 168, 192, 216, and 240
Population: TIO analysis set with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Burosumab
Number analyzed (Participants) | 14
pg/mL
  Week 24 | 246335.35 (61089.98)
  Week 48: number analyzed (Participants) | 10
  Week 48 | 180511.74 (33529.14)
  Week 96: number analyzed (Participants) | 11
  Week 96 | 331267.40 (103226.37)
  Week 144: number analyzed (Participants) | 11
  Week 144 | 275758.40 (102349.79)
  Week 168: number analyzed (Participants) | 10
  Week 168 | 185769.23 (65423.93)
  Week 192: number analyzed (Participants) | 9
  Week 192 | 234826.20 (82198.24)
  Week 216: number analyzed (Participants) | 7
  Week 216 | 254359.96 (81615.67)
  Week 240: number analyzed (Participants) | 7
  Week 240 | 210119.10 (76610.50)
Statistical Analysis 1: Comparison: Burosumab; Week 24; Test type: Other; p < 0.0001, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline total FGF23
Statistical Analysis 2: Comparison: Burosumab; Week 48; Test type: Other; p < 0.0001, GEE model; [statistical method as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: Burosumab; Week 96; Test type: Other; p = 0.001, GEE model; [statistical method as in outcome 13, analysis 1]
Statistical Analysis 4: Comparison: Burosumab; Week 144; Test type: Other; p = 0.007, GEE model; [statistical method as in outcome 13, analysis 1]
Statistical Analysis 5: Comparison: Burosumab; Week 168; Test type: Other; p = 0.005, GEE model; [statistical method as in outcome 13, analysis 1]
Statistical Analysis 6: Comparison: Burosumab; Week 192; Test type: Other; p = 0.004, GEE model; [statistical method as in outcome 13, analysis 1]
Statistical Analysis 7: Comparison: Burosumab; Week 216; Test type: Other; p = 0.002, GEE model; [statistical method as in outcome 13, analysis 1]
Statistical Analysis 8: Comparison: Burosumab; Week 240; Test type: Other; p = 0.006, GEE model; [statistical method as in outcome 13, analysis 1]

14. Secondary Outcome: Change From Baseline Over Time in Free Serum Fibroblast Growth Factor 23 (FGF23) Concentration
Description: Least squares means and standard errors were estimated from a generalized estimation equation (GEE) model which includes the change from Baseline as the dependent variable, time as the categorical variable and adjusted for Baseline free FGF23, with compound symmetry covariance structure.
Time Frame: Baseline and Weeks 24, 48, 96, 144, 168, 192, 216, and 240
Population: TIO analysis set with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Burosumab
Number analyzed (Participants) | 14
pg/mL
  Week 24 | 624.91 (101.89)
  Week 48: number analyzed (Participants) | 11
  Week 48 | 578.07 (95.37)
  Week 96: number analyzed (Participants) | 12
  Week 96 | 736.59 (139.18)
  Week 144: number analyzed (Participants) | 11
  Week 144 | 801.69 (103.41)
  Week 168: number analyzed (Participants) | 10
  Week 168 | 787.16 (95.52)
  Week 192: number analyzed (Participants) | 9
  Week 192 | 717.71 (115.99)
  Week 216: number analyzed (Participants) | 7
  Week 216 | 704.87 (115.30)
  Week 240: number analyzed (Participants) | 7
  Week 240 | 625.16 (125.93)
Statistical Analysis 1: Comparison: Burosumab; Week 24; Test type: Other; p < 0.001, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline free FGF23
Statistical Analysis 2: Comparison: Burosumab; Week 48; Test type: Other; p < 0.001, GEE model; [statistical method as in outcome 14, analysis 1]
Statistical Analysis 3: Comparison: Burosumab; Week 96; Test type: Other; p < 0.001, GEE model; [statistical method as in outcome 14, analysis 1]
Statistical Analysis 4: Comparison: Burosumab; Week 144; Test type: Other; p < 0.001, GEE model; [statistical method as in outcome 14, analysis 1]
Statistical Analysis 5: Comparison: Burosumab; Week 168; Test type: Other; p < 0.001, GEE model; [statistical method as in outcome 14, analysis 1]
Statistical Analysis 6: Comparison: Burosumab; Week 192; Test type: Other; p < 0.001, GEE model; [statistical method as in outcome 14, analysis 1]
Statistical Analysis 7: Comparison: Burosumab; Week 216; Test type: Other; p < 0.001, GEE model; [statistical method as in outcome 14, analysis 1]
Statistical Analysis 8: Comparison: Burosumab; Week 240; Test type: Other; p < 0.001, GEE model; [statistical method as in outcome 14, analysis 1]

15. Secondary Outcome: Change From Baseline Over Time in 24-hour Urinary Phosphorus
Description: Least squares means and standard errors were estimated from a generalized estimation equation (GEE) model which includes the change from Baseline as the dependent variable, time as the categorical variable and adjusted for Baseline 24-hour urinary phosphorus, with compound symmetry covariance structure.
Time Frame: Baseline and Weeks 24, 48, 96, 144, 168, 192, 216, and 240
Population: TIO analysis set participants with available data at each time point.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Burosumab
Number analyzed (Participants) | 14
mg/dL
  Week 24: number analyzed (Participants) | 11
  Week 24 | -3.66 (8.28)
  Week 48: number analyzed (Participants) | 13
  Week 48 | 3.59 (6.73)
  Week 96: number analyzed (Participants) | 9
  Week 96 | 3.22 (6.40)
  Week 144: number analyzed (Participants) | 8
  Week 144 | 3.25 (6.971)
  Week 168: number analyzed (Participants) | 10
  Week 168 | 4.98 (8.18)
  Week 192: number analyzed (Participants) | 8
  Week 192 | 8.31 (4.54)
  Week 216: number analyzed (Participants) | 7
  Week 216 | 13.93 (14.30)
  Week 240: number analyzed (Participants) | 6
  Week 240 | 13.11 (9.35)
Statistical Analysis 1: Comparison: Burosumab; Week 24; Test type: Other; p = 0.659, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline 24-hour urinary phosphorus
Statistical Analysis 2: Comparison: Burosumab; Week 48; Test type: Other; p = 0.752, GEE model; [statistical method as in outcome 15, analysis 1]
Statistical Analysis 3: Comparison: Burosumab; Week 96; Test type: Other; p = 0.594, GEE model; [statistical method as in outcome 15, analysis 1]
Statistical Analysis 4: Comparison: Burosumab; Week 144; Test type: Other; p = 0.614, GEE model; [statistical method as in outcome 15, analysis 1]
Statistical Analysis 5: Comparison: Burosumab; Week 168; Test type: Other; p = 0.542, GEE model; [statistical method as in outcome 15, analysis 1]
Statistical Analysis 6: Comparison: Burosumab; Week 192; Test type: Other; p = 0.067, GEE model; [statistical method as in outcome 15, analysis 1]
Statistical Analysis 7: Comparison: Burosumab; Week 216; Test type: Other; p = 0.330, GEE model; [statistical method as in outcome 15, analysis 1]
Statistical Analysis 8: Comparison: Burosumab; Week 240; Test type: Superiority; p = 0.161, GEE model; [statistical method as in outcome 15, analysis 1]

16. Secondary Outcome: Change From Baseline Over Time in Tubular Reabsorption of Phosphate (TRP)
Description: Tubular reabsorption of phosphate (TRP) is the fraction of filtered phosphorus that is reabsorbed by renal tubules.
  Least squares means and standard errors were estimated from a generalized estimation equation (GEE) model which includes the change from Baseline as the dependent variable, time as the categorical variable and adjusted for Baseline TRP, with compound symmetry covariance structure.
Time Frame: Baseline and Weeks 24, 48, 96, 144, 168, 192, 216, and 240
Population: TIO analysis set participants with available data at Baseline and each time point.
Measure: Least Squares Mean (Standard Error); unit: fraction of phosphorus reabsorbed
Arm/Group | Burosumab
Number analyzed (Participants) | 13
fraction of phosphorus reabsorbed
  Week 24: number analyzed (Participants) | 12
  Week 24 | 0.13 (0.02)
  Week 48: number analyzed (Participants) | 12
  Week 48 | 0.14 (0.02)
  Week 96: number analyzed (Participants) | 11
  Week 96 | 0.10 (0.03)
  Week 144: number analyzed (Participants) | 9
  Week 144 | 0.13 (0.02)
  Week 168: number analyzed (Participants) | 9
  Week 168 | 0.12 (0.02)
  Week 192: number analyzed (Participants) | 7
  Week 192 | 0.14 (0.02)
  Week 216: number analyzed (Participants) | 6
  Week 216 | 0.14 (0.01)
  Week 240: number analyzed (Participants) | 6
  Week 240 | 0.12 (0.02)
Statistical Analysis 1: Comparison: Burosumab; Week 24; Test type: Other; p < 0.001, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline TRP
Statistical Analysis 2: Comparison: Burosumab; Week 48; Test type: Other; p < 0.001, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline TRP
Statistical Analysis 3: Comparison: Burosumab; Week 96; Test type: Other; p = 0.001, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline TRP
Statistical Analysis 4: Comparison: Burosumab; Week 144; Test type: Other; p < 0.001, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline TRP
Statistical Analysis 5: Comparison: Burosumab; Week 168; Test type: Other; p < 0.001, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline TRP
Statistical Analysis 6: Comparison: Burosumab; Week 192; Test type: Superiority; p < 0.001, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline TRP
Statistical Analysis 7: Comparison: Burosumab; Week 216; Test type: Superiority; p < 0.001, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline TRP
Statistical Analysis 8: Comparison: Burosumab; Week 240; Test type: Superiority; p < 0.001, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline TRP

17. Secondary Outcome: Change From Baseline Over Time in Ratio of Renal Tubular Maximum Phosphate Reabsorption Rate to Glomerular Filtration Rate (TmP/GFR)
Description: TmP/GFR measures renal phosphate reabsorption (the primary mechanism by which FGF23 regulates phosphate homeostasis) by comparing the fractional absorption of phosphate relative to the estimated rate of glomerular filtration.
  Least squares means and standard errors were estimated from a generalized estimation equation (GEE) model which includes the change from Baseline as the dependent variable, time as the categorical variable and adjusted for Baseline TmP/GFR, with compound symmetry covariance structure.
Time Frame: Baseline and Weeks 24, 48, 96, 144, 168, 192, 216, and 240
Population: TIO analysis set participants with available data at Baseline and each time point.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Burosumab
Number analyzed (Participants) | 13
mg/dL
  Week 24: number analyzed (Participants) | 12
  Week 24 | 0.81 (0.13)
  Week 48: number analyzed (Participants) | 12
  Week 48 | 0.88 (0.14)
  Week 96: number analyzed (Participants) | 11
  Week 96 | 0.73 (0.23)
  Week 144: number analyzed (Participants) | 9
  Week 144 | 0.13 (0.02)
  Week 168: number analyzed (Participants) | 9
  Week 168 | 1.07 (0.29)
  Week 192: number analyzed (Participants) | 7
  Week 192 | 0.95 (0.16)
  Week 216: number analyzed (Participants) | 6
  Week 216 | 0.88 (0.12)
  Week 240: number analyzed (Participants) | 6
  Week 240 | 0.94 (0.15)
Statistical Analysis 1: Comparison: Burosumab; Week 24; Test type: Other; p < 0.001, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline TmP/GFR
Statistical Analysis 2: Comparison: Burosumab; Week 48; Test type: Other; p < 0.001, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline TmP/GFR
Statistical Analysis 3: Comparison: Burosumab; Week 96; Test type: Other; p = 0.002, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline TmP/GFR
Statistical Analysis 4: Comparison: Burosumab; Week 144; Test type: Other; p < 0.001, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline TmP/GFR
Statistical Analysis 5: Comparison: Burosumab; Week 168; Test type: Other; p < 0.001, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline TmP/GFR
Statistical Analysis 6: Comparison: Burosumab; Week 192; Test type: Other; p < 0.001, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline TmP/GFR
Statistical Analysis 7: Comparison: Burosumab; Week 216; Test type: Other; p < 0.001, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline TmP/GFR
Statistical Analysis 8: Comparison: Burosumab; Week 240; Test type: Other; p < 0.001, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline TmP/GFR

18. Secondary Outcome: Change From Baseline Over Time in Fractional Excretion of Phosphorus (FEP)
Description: FEP is the percentage of phosphorus filtered by the kidney that is excreted into urine, calculated as 100% * (2-hour urine phosphorus*serum creatinine)/(2-hour urine creatinine * serum phosphorus).
  Least squares means and standard errors were estimated from a generalized estimation equation (GEE) model which includes the change from Baseline as the dependent variable, time as the categorical variable and adjusted for Baseline FEP, with compound symmetry covariance structure.
Time Frame: Baseline and Weeks 24, 48, 96, 144, 168, 192, 216, and 240
Population: TIO analysis set participants with available data at each time point.
Measure: Least Squares Mean (Standard Error); unit: percentage of phosphorus
Arm/Group | Burosumab
Number analyzed (Participants) | 14
percentage of phosphorus
  Week 24 | -0.14 (0.02)
  Week 48: number analyzed (Participants) | 13
  Week 48 | -0.14 (0.02)
  Week 96: number analyzed (Participants) | 12
  Week 96 | -0.10 (0.03)
  Week 144: number analyzed (Participants) | 10
  Week 144 | -0.15 (0.02)
  Week 168: number analyzed (Participants) | 10
  Week 168 | -0.14 (0.02)
  Week 192: number analyzed (Participants) | 8
  Week 192 | -0.14 (0.02)
  Week 216: number analyzed (Participants) | 7
  Week 216 | -0.15 (0.01)
  Week 240: number analyzed (Participants) | 7
  Week 240 | -0.14 (0.02)
Statistical Analysis 1: Comparison: Burosumab; Week 24; Test type: Other; p < 0.001, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline FEP
Statistical Analysis 2: Comparison: Burosumab; Week 48; Test type: Other; p < 0.001, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline FEP
Statistical Analysis 3: Comparison: Burosumab; Week 96; Test type: Other; p < 0.001, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline FEP
Statistical Analysis 4: Comparison: Burosumab; Week 144; Test type: Other; p < 0.001, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline FEP
Statistical Analysis 5: Comparison: Burosumab; Week 168; Test type: Other; p < 0.001, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline FEP
Statistical Analysis 6: Comparison: Burosumab; Week 192; Test type: Other; p < 0.001, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline FEP
Statistical Analysis 7: Comparison: Burosumab; Week 216; Test type: Other; p < 0.001, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline FEP
Statistical Analysis 8: Comparison: Burosumab; Week 240; Test type: Other; p < 0.001, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline FEP

19. Secondary Outcome: Change From Baseline Over Time in Serum Alkaline Phosphatase (ALP)
Description: Least squares means and standard errors were estimated from a generalized estimation equation (GEE) model which includes the change from Baseline as the dependent variable, time as the categorical variable and adjusted for Baseline ALP, with compound symmetry covariance structure.
Time Frame: Baseline and Weeks 24, 48, 96, 144, 168, 192, 216, and 240
Population: TIO analysis set participants with available data at each time point.
Measure: Least Squares Mean (Standard Error); unit: U/L
Arm/Group | Burosumab
Number analyzed (Participants) | 14
U/L
  Week 24 | -1.68 (10.91)
  Week 48: number analyzed (Participants) | 13
  Week 48 | -20.36 (11.68)
  Week 96: number analyzed (Participants) | 12
  Week 96 | -38.23 (11.90)
  Week 144: number analyzed (Participants) | 11
  Week 144 | -57.45 (10.97)
  Week 168: number analyzed (Participants) | 10
  Week 168 | -62.80 (12.35)
  Week 192: number analyzed (Participants) | 10
  Week 192 | -60.40 (12.41)
  Week 216: number analyzed (Participants) | 7
  Week 216 | -50.14 (26.09)
  Week 240: number analyzed (Participants) | 7
  Week 240 | -49.71 (24.35)
Statistical Analysis 1: Comparison: Burosumab; Week 24; Test type: Other; p = 0.878, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline ALP
Statistical Analysis 2: Comparison: Burosumab; Week 48; Test type: Other; p = 0.081, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline ALP
Statistical Analysis 3: Comparison: Burosumab; Week 96; Test type: Other; p = 0.001, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline ALP
Statistical Analysis 4: Comparison: Burosumab; Week 144; Test type: Other; p < 0.001, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline ALP
Statistical Analysis 5: Comparison: Burosumab; Week 168; Test type: Other; p < 0.001, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline ALP
Statistical Analysis 6: Comparison: Burosumab; Week 192; Test type: Other; p < 0.001, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline ALP
Statistical Analysis 7: Comparison: Burosumab; Week 216; Test type: Other; p = 0.055, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline ALP
Statistical Analysis 8: Comparison: Burosumab; Week 240; Test type: Other; p = 0.041, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline ALP

20. Secondary Outcome: Change From Baseline Over Time in Bone-Specific Alkaline Phosphatase (BALP)
Description: Least squares means and standard errors were estimated from a generalized estimation equation (GEE) model which includes the change from Baseline as the dependent variable, time as the categorical variable and adjusted for Baseline BALP, with compound symmetry covariance structure.
Time Frame: Baseline and Weeks 24, 48, 96, 144, 168, 192, 216, and 240
Population: TIO analysis set participants with available data at each time point.
Measure: Least Squares Mean (Standard Error); unit: μg/L
Arm/Group | Burosumab
Number analyzed (Participants) | 14
μg/L
  Week 24 | -1.13 (4.87)
  Week 48: number analyzed (Participants) | 12
  Week 48 | -9.65 (4.74)
  Week 96: number analyzed (Participants) | 12
  Week 96 | -15.89 (4.27)
  Week 144: number analyzed (Participants) | 11
  Week 144 | -19.81 (4.42)
  Week 168: number analyzed (Participants) | 10
  Week 168 | -22.05 (4.52)
  Week 192: number analyzed (Participants) | 10
  Week 192 | -21.54 (4.87)
  Week 216: number analyzed (Participants) | 7
  Week 216 | -15.50 (11.39)
  Week 240: number analyzed (Participants) | 7
  Week 240 | -21.58 (6.17)
Statistical Analysis 1: Comparison: Burosumab; Week 24; Test type: Other; p = 0.817, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline BALP
Statistical Analysis 2: Comparison: Burosumab; Week 48; Test type: Other; p = 0.042, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline BALP
Statistical Analysis 3: Comparison: Burosumab; Week 96; Test type: Other; p < 0.001, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline BALP
Statistical Analysis 4: Comparison: Burosumab; Week 144; Test type: Other; p < 0.001, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline BALP
Statistical Analysis 5: Comparison: Burosumab; Week 168; Test type: Other; p < 0.001, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline BALP
Statistical Analysis 6: Comparison: Burosumab; Week 192; Test type: Other; p < 0.001, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline BALP
Statistical Analysis 7: Comparison: Burosumab; Week 216; Test type: Other; p = 0.174, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline BALP
Statistical Analysis 8: Comparison: Burosumab; Week 240; Test type: Other; p < 0.001, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline BALP

21. Secondary Outcome: Percent Change From Baseline Over Time in BALP
Description: as for outcome 20
Time Frame: Baseline and Weeks 24, 48, 96, 144, 168, 192, 216, and 240
Population: TIO analysis set participants with available data at each time point.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Burosumab
Number analyzed (Participants) | 14
percent change
  Week 24 | 5.15 (13.06)
  Week 48: number analyzed (Participants) | 12
  Week 48 | -16.56 (8.35)
  Week 96: number analyzed (Participants) | 12
  Week 96 | -30.40 (8.57)
  Week 144: number analyzed (Participants) | 11
  Week 144 | -35.82 (9.47)
  Week 168: number analyzed (Participants) | 10
  Week 168 | -40.97 (9.60)
  Week 192: number analyzed (Participants) | 10
  Week 192 | -41.11 (9.93)
  Week 216: number analyzed (Participants) | 7
  Week 216 | -28.41 (20.71)
  Week 240: number analyzed (Participants) | 7
  Week 240 | -42.27 (11.65)
Statistical Analysis 1: Comparison: Burosumab; Week 24; Test type: Other; p = 0.694, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline BALP
Statistical Analysis 2: Comparison: Burosumab; Week 48; Test type: Other; p = 0.047, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline BALP
Statistical Analysis 3: Comparison: Burosumab; Week 96; Test type: Other; p < 0.001, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline BALP
Statistical Analysis 4: Comparison: Burosumab; Week 144; Test type: Other; p < 0.001, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline BALP
Statistical Analysis 5: Comparison: Burosumab; Week 168; Test type: Other; p < 0.001, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline BALP
Statistical Analysis 6: Comparison: Burosumab; Week 192; Test type: Other; p < 0.001, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline BALP
Statistical Analysis 7: Comparison: Burosumab; Week 216; Test type: Other; p = 0.170, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline BALP
Statistical Analysis 8: Comparison: Burosumab; Week 240; Test type: Other; p < 0.001, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline BALP

22. Secondary Outcome: Change From Baseline Over Time in Carboxy Terminal Cross-Linked Telopeptide of Type 1 Collagen (CTx)
Description: Least squares means and standard errors were estimated from a generalized estimation equation (GEE) model which includes the change from Baseline as the dependent variable, time as the categorical variable and adjusted for Baseline CTx, with compound symmetry covariance structure.
Time Frame: Baseline and Weeks 24, 48, 96, 144, 168, 192, 216, and 240
Population: TIO analysis set participants with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Burosumab
Number analyzed (Participants) | 14
pg/mL
  Week 24 | 212.91 (125.76)
  Week 48: number analyzed (Participants) | 13
  Week 48 | 97.02 (80.10)
  Week 96: number analyzed (Participants) | 12
  Week 96 | 6.55 (63.66)
  Week 144: number analyzed (Participants) | 11
  Week 144 | -19.28 (38.49)
  Week 168: number analyzed (Participants) | 10
  Week 168 | -100.84 (49.31)
  Week 192: number analyzed (Participants) | 9
  Week 192 | -200.40 (65.80)
  Week 216: number analyzed (Participants) | 7
  Week 216 | -140.71 (94.55)
  Week 240: number analyzed (Participants) | 7
  Week 240 | -92.14 (102.27)
Statistical Analysis 1: Comparison: Burosumab; Week 24; Test type: Other; p = 0.090, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline CTx
Statistical Analysis 2: Comparison: Burosumab; Week 48; Test type: Other; p = 0.226, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline CTx
Statistical Analysis 3: Comparison: Burosumab; Week 96; Test type: Other; p = 0.918, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline CTx
Statistical Analysis 4: Comparison: Burosumab; Week 144; Test type: Other; p = 0.616, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline CTx
Statistical Analysis 5: Comparison: Burosumab; Week 168; Test type: Other; p = 0.041, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline CTx
Statistical Analysis 6: Comparison: Burosumab; Week 192; Test type: Other; p = 0.002, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline CTx
Statistical Analysis 7: Comparison: Burosumab; Week 216; Test type: Other; p = 0.137, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline CTx
Statistical Analysis 8: Comparison: Burosumab; Week 240; Test type: Other; p = 0.368, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline CTx

23. Secondary Outcome: Percent Change From Baseline Over Time in CTx
Description: as for outcome 22
Time Frame: Baseline and Weeks 24, 48, 96, 144, 168, 192, 216, and 240
Population: TIO analysis set participants with available data at each time point.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Burosumab
Number analyzed (Participants) | 14
percent change
  Week 24 | 33.77 (14.33)
  Week 48: number analyzed (Participants) | 13
  Week 48 | 31.05 (20.220)
  Week 96: number analyzed (Participants) | 12
  Week 96 | 11.96 (12.05)
  Week 144: number analyzed (Participants) | 11
  Week 144 | 10.92 (8.86)
  Week 168: number analyzed (Participants) | 10
  Week 168 | -2.23 (8.29)
  Week 192: number analyzed (Participants) | 9
  Week 192 | -15.90 (11.21)
  Week 216: number analyzed (Participants) | 7
  Week 216 | -10.53 (7.40)
  Week 240: number analyzed (Participants) | 7
  Week 240 | -5.68 (10.26)
Statistical Analysis 1: Comparison: Burosumab; Week 24; Test type: Other; p = 0.018, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline CTx
Statistical Analysis 2: Comparison: Burosumab; Week 48; Test type: Other; p = 0.133, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline CTx
Statistical Analysis 3: Comparison: Burosumab; Week 96; Test type: Other; p = 0.321, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline CTx
Statistical Analysis 4: Comparison: Burosumab; Week 144; Test type: Other; p = 0.218, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline CTx
Statistical Analysis 5: Comparison: Burosumab; Week 168; Test type: Other; p = 0.788, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline CTx
Statistical Analysis 6: Comparison: Burosumab; Week 192; Test type: Other; p = 0.156, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline CTx
Statistical Analysis 7: Comparison: Burosumab; Week 216; Test type: Other; p = 0.155, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline CTx
Statistical Analysis 8: Comparison: Burosumab; Week 240; Test type: Other; p = 0.580, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline CTx

24. Secondary Outcome: Change From Baseline Over Time in Procollagen Type 1 N-Propeptide (P1NP)
Description: Least squares means and standard errors were estimated from a generalized estimation equation (GEE) model which includes the change from Baseline as the dependent variable, time as the categorical variable and adjusted for Baseline P1NP, with compound symmetry covariance structure.
Time Frame: Baseline and Weeks 24, 48, 96, 144, 168, 192, 216, and 240
Population: TIO analysis set participants with available data at each time point.
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Burosumab
Number analyzed (Participants) | 14
ng/mL
  Week 24 | 34.07 (10.90)
  Week 48: number analyzed (Participants) | 13
  Week 48 | 7.73 (7.05)
  Week 96: number analyzed (Participants) | 12
  Week 96 | 11.28 (15.56)
  Week 144: number analyzed (Participants) | 11
  Week 144 | 1.21 (5.55)
  Week 168: number analyzed (Participants) | 9
  Week 168 | -12.04 (3.36)
  Week 192: number analyzed (Participants) | 10
  Week 192 | -11.93 (8.11)
  Week 216: number analyzed (Participants) | 7
  Week 216 | -7.53 (14.58)
  Week 240: number analyzed (Participants) | 7
  Week 240 | -1.67 (14.39)
Statistical Analysis 1: Comparison: Burosumab; Week 24; Test type: Other; p = 0.002, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline P1NP
Statistical Analysis 2: Comparison: Burosumab; Week 48; Test type: Other; p = 0.273, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline P1NP
Statistical Analysis 3: Comparison: Burosumab; Week 96; Test type: Other; p = 0.469, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline P1NP
Statistical Analysis 4: Comparison: Burosumab; Week 144; Test type: Other; p = 0.828, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline P1NP
Statistical Analysis 5: Comparison: Burosumab; Week 168; Test type: Other; p < 0.001, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline P1NP
Statistical Analysis 6: Comparison: Burosumab; Week 192; Test type: Other; p = 0.141, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline P1NP
Statistical Analysis 7: Comparison: Burosumab; Week 216; Test type: Other; p = 0.606, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline P1NP
Statistical Analysis 8: Comparison: Burosumab; Week 240; Test type: Other; p = 0.907, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline P1NP

25. Secondary Outcome: Percent Change From Baseline Over Time in P1NP
Description: as for outcome 24
Time Frame: Baseline and Weeks 24, 48, 96, 144, 168, 192, 216, and 240
Population: TIO analysis set participants with available data at each time point.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Burosumab
Number analyzed (Participants) | 14
percent change
  Week 24 | 53.71 (16.35)
  Week 48: number analyzed (Participants) | 13
  Week 48 | 15.64 (10.84)
  Week 96: number analyzed (Participants) | 12
  Week 96 | 18.09 (20.29)
  Week 144: number analyzed (Participants) | 11
  Week 144 | 13.65 (8.68)
  Week 168: number analyzed (Participants) | 9
  Week 168 | -12.40 (4.98)
  Week 192: number analyzed (Participants) | 10
  Week 192 | 0.93 (19.78)
  Week 216: number analyzed (Participants) | 7
  Week 216 | -7.58 (17.45)
  Week 240: number analyzed (Participants) | 7
  Week 240 | 4.47 (16.82)
Statistical Analysis 1: Comparison: Burosumab; Week 24; Test type: Other; p = 0.001, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline P1NP
Statistical Analysis 2: Comparison: Burosumab; Week 48; Test type: Other; p = 0.149, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline P1NP
Statistical Analysis 3: Comparison: Burosumab; Week 96; Test type: Other; p = 0.372, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline P1NP
Statistical Analysis 4: Comparison: Burosumab; Week 144; Test type: Other; p = 0.116, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline P1NP
Statistical Analysis 5: Comparison: Burosumab; Week 168; Test type: Other; p = 0.013, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline P1NP
Statistical Analysis 6: Comparison: Burosumab; Week 192; Test type: Other; p = 0.962, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline P1NP
Statistical Analysis 7: Comparison: Burosumab; Week 216; Test type: Other; p = 0.664, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline P1NP
Statistical Analysis 8: Comparison: Burosumab; Week 240; Test type: Other; p = 0.790, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline P1NP

26. Secondary Outcome: Change From Baseline Over Time in Osteocalcin
Description: Least squares means and standard errors were estimated from a generalized estimation equation (GEE) model which includes the change from Baseline as the dependent variable, time as the categorical variable and adjusted for Baseline osteocalcin, with compound symmetry covariance structure.
Time Frame: Baseline and Weeks 24, 48, 96, 144, 168, 192, 216, and 240
Population: TIO analysis set with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Burosumab
Number analyzed (Participants) | 14
ng/mL
  Week 24 | 9.51 (4.85)
  Week 48: number analyzed (Participants) | 11
  Week 48 | 2.20 (3.48)
  Week 96: number analyzed (Participants) | 12
  Week 96 | -0.54 (2.75)
  Week 144: number analyzed (Participants) | 10
  Week 144 | -0.52 (1.89)
  Week 168: number analyzed (Participants) | 10
  Week 168 | -3.14 (1.35)
  Week 192: number analyzed (Participants) | 10
  Week 192 | -6.91 (2.49)
  Week 216: number analyzed (Participants) | 6
  Week 216 | -7.97 (5.35)
  Week 240: number analyzed (Participants) | 7
  Week 240 | -8.55 (5.22)
Statistical Analysis 1: Comparison: Burosumab; Week 24; Test type: Other; p = 0.050, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline osteocalcin
Statistical Analysis 2: Comparison: Burosumab; Week 48; Test type: Other; p = 0.526, GEE model; [statistical method as in outcome 26, analysis 1]
Statistical Analysis 3: Comparison: Burosumab; Week 96; Test type: Other; p = 0.845, GEE model; [statistical method as in outcome 26, analysis 1]
Statistical Analysis 4: Comparison: Burosumab; Week 144; Test type: Other; p = 0.782, GEE model; [statistical method as in outcome 26, analysis 1]
Statistical Analysis 5: Comparison: Burosumab; Week 168; Test type: Other; p = 0.020, GEE model; [statistical method as in outcome 26, analysis 1]
Statistical Analysis 6: Comparison: Burosumab; Week 192; Test type: Other; p = 0.005, GEE model; [statistical method as in outcome 26, analysis 1]
Statistical Analysis 7: Comparison: Burosumab; Week 216; Test type: Other; p = 0.136, GEE model; [statistical method as in outcome 26, analysis 1]
Statistical Analysis 8: Comparison: Burosumab; Week 240; Test type: Other; p = 0.101, GEE model; [statistical method as in outcome 26, analysis 1]

27. Secondary Outcome: Percent Change From Baseline Over Time in Osteocalcin
Description: as for outcome 26
Time Frame: Baseline and Weeks 24, 48, 96, 144, 168, 192, 216, and 240
Population: TIO analysis set with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Burosumab
Number analyzed (Participants) | 14
percent change
  Week 24 | 41.49 (12.19)
  Week 48: number analyzed (Participants) | 11
  Week 48 | 16.28 (13.79)
  Week 96: number analyzed (Participants) | 12
  Week 96 | 15.04 (14.10)
  Week 144: number analyzed (Participants) | 10
  Week 144 | 14.08 (8.38)
  Week 168: number analyzed (Participants) | 10
  Week 168 | -0.98 (7.11)
  Week 192: number analyzed (Participants) | 10
  Week 192 | -19.67 (10.42)
  Week 216: number analyzed (Participants) | 6
  Week 216 | -5.65 (11.48)
  Week 240: number analyzed (Participants) | 7
  Week 240 | -8.37 (10.17)
Statistical Analysis 1: Comparison: Burosumab; Week 24; Test type: Other; p < 0.001, GEE model; [statistical method as in outcome 26, analysis 1]
Statistical Analysis 2: Comparison: Burosumab; Week 48; Test type: Other; p = 0.238, GEE model; [statistical method as in outcome 26, analysis 1]
Statistical Analysis 3: Comparison: Burosumab; Week 96; Test type: Other; p = 0.286, GEE model; [statistical method as in outcome 26, analysis 1]
Statistical Analysis 4: Comparison: Burosumab; Week 144; Test type: Other; p = 0.093, GEE model; [statistical method as in outcome 26, analysis 1]
Statistical Analysis 5: Comparison: Burosumab; Week 168; Test type: Other; p = 0.890, GEE model; [statistical method as in outcome 26, analysis 1]
Statistical Analysis 6: Comparison: Burosumab; Week 192; Test type: Other; p = 0.059, GEE model; [statistical method as in outcome 26, analysis 1]
Statistical Analysis 7: Comparison: Burosumab; Week 216; Test type: Superiority; p = 0.623, GEE model — Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline osteocalcin
Statistical Analysis 8: Comparison: Burosumab; Week 240; Test type: Other; p = 0.411, GEE model; [statistical method as in outcome 26, analysis 1]

28. Secondary Outcome: Change From Baseline Over Time in Hand-Held Dynamometry (HHD) Elbow Measurements
Description: To assess muscle strength, hand-held dynamometry was conducted using a standardized technique. Bilateral strength (defined as the average of the left and the right scores, measured in kilograms) of the elbow flexors and extensors was measured by the maximum voluntary isometric contraction against a dynamometer.
  Least squares means and standard errors were estimated from a generalized estimation equation (GEE) model which includes the change from Baseline as the dependent variable, time as the categorical variable and adjusted for Baseline strength measurements, with compound symmetry covariance structure.
Time Frame: Baseline and Weeks 24 and 48
Population: TIO analysis set with available elbow dynamometry measurements at Baseline and each time point.
Measure: Least Squares Mean (Standard Error); unit: kg
Groups:
- Elbow Flexion: Elbow flexor (biceps brachii, brachioradialis, and brachialis) muscle strength was measured in participants who received burosumab at a starting dose of 0.3 mg/kg administered subcutaneously Q4W. Doses may have been titrated up to a maximum of 2.0 mg/kg Q2W.
- Elbow Extension: Elbow extensor (triceps brachii and anconeus) muscle strength was measured in participants who received burosumab at a starting dose of 0.3 mg/kg administered subcutaneously Q4W. Doses may have been titrated up to a maximum of 2.0 mg/kg Q2W.
Arm/Group | Elbow Flexion | Elbow Extension
Number analyzed (Participants) | 9 | 9
kg
  Week 24: number analyzed (Participants) | 8 | 8
  Week 24 | 0.12 (0.512) | 0.75 (0.704)
  Week 48: number analyzed (Participants) | 8 | 8
  Week 48 | 0.32 (0.753) | 1.06 (0.760)
Statistical Analysis 1: Comparison: Elbow Flexion; Week 24; Test type: Other; p = 0.8209, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline measurement
Statistical Analysis 2: Comparison: Elbow Extension; Week 24; Test type: Other; p = 0.2851, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 3: Comparison: Elbow Flexion; Week 48; Test type: Other; p = 0.6689, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 4: Comparison: Elbow Extension; Week 48; Test type: Other; p = 0.1612, GEE model; [statistical method as in outcome 28, analysis 1]

29. Secondary Outcome: Change From Baseline Over Time in Hand-Held Dynamometry (HHD) Knee Measurements
Description: To assess muscle strength, hand-held dynamometry was conducted using a standardized technique. Bilateral strength (defined as the average of the left and the right scores, measured in kilograms) of the knee flexors and extensors was measured by the maximum voluntary isometric contraction against a dynamometer.
  Least squares means and standard errors were estimated from a generalized estimation equation (GEE) model which includes the change from Baseline as the dependent variable, time as the categorical variable and adjusted for Baseline strength measurements, with compound symmetry covariance structure.
Time Frame: Baseline and Weeks 24 and 48
Population: TIO analysis set with available knee dynamometry measurements at Baseline and each time point.
Measure: Least Squares Mean (Standard Error); unit: kg
Groups:
- Knee Flexion: Knee flexor (hamstring) muscle strength was measured in participants who received burosumab at a starting dose of 0.3 mg/kg administered subcutaneously Q4W. Doses may have been titrated up to a maximum of 2.0 mg/kg Q2W.
- Knee Extension: Knee extensor (quadriceps) muscle strength was measured in participants who received burosumab at a starting dose of 0.3 mg/kg administered subcutaneously Q4W. Doses may have been titrated up to a maximum of 2.0 mg/kg Q2W.
Arm/Group | Knee Flexion | Knee Extension
Number analyzed (Participants) | 10 | 10
kg
  Week 24: number analyzed (Participants) | 9 | 9
  Week 24 | 0.94 (1.139) | -0.89 (1.573)
  Week 48: number analyzed (Participants) | 9 | 9
  Week 48 | 1.21 (1.297) | 0.75 (1.158)
Statistical Analysis 1: Comparison: Knee Flexion; Week 24; Test type: Other; p = 0.4093, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 2: Comparison: Knee Extension; Week 24; Test type: Other; p = 0.5720, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 3: Comparison: Knee Flexion; Week 48; Test type: Other; p = 0.3501, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 4: Comparison: Knee Extension; Week 48; Test type: Other; p = 0.5172, GEE model; [statistical method as in outcome 28, analysis 1]

30. Secondary Outcome: Change From Baseline Over Time in Sit-to-Stand (STS) Test
Description: The STS test measures lower extremity strength and mobility as a participant moves repeatedly from a seated position to standing. This study used a modified STS test that allowed participants to use the arms of the chair to help them stand and sit if necessary. The number of sit-to-stand repetitions performed in a 30-second period was recorded.
  Least squares means and standard errors were estimated from a generalized estimation equation (GEE) model which includes the change from Baseline as the dependent variable, time as the categorical variable and adjusted for Baseline measurement, with compound symmetry covariance structure.
Time Frame: Baseline and Weeks 24 and 48
Population: TIO analysis set with available STS data at each time point; One participant did not perform the test at Baseline as it was not included in the original protocol, and 2 participants were unable to perform the test due to underlying medical issues.
Measure: Least Squares Mean (Standard Error); unit: sit-to-stand repetitions
Arm/Group | Burosumab
Number analyzed (Participants) | 11
sit-to-stand repetitions
  Week 24: number analyzed (Participants) | 10
  Week 24 | 1.5 (0.54)
  Week 48: number analyzed (Participants) | 10
  Week 48 | 1.6 (0.50)
Statistical Analysis 1: Comparison: Burosumab; Week 24; Test type: Other; p = 0.0046, GEE model; Generalized estimation equation (GEE) model includes time as the categorical variable and adjusted for Baseline STS measurement
Statistical Analysis 2: Comparison: Burosumab; Week 48; Test type: Other; p = 0.0012, GEE model; [statistical method as in outcome 30, analysis 1]

31. Secondary Outcome: Change From Baseline Over Time in Weighted Arm Lift (WAL) Test
Description: The Weighted arm lift (WAL) test assesses upper extremity strength, mobility and reaching ability. The test was administered bilaterally to determine the number of times the participant could raise a 1 kg weight above the head in a 30-second period. The number of repetitions completed with each arm was recorded.
  Least squares means and standard errors were estimated from a generalized estimation equation (GEE) model which includes the change from Baseline as the dependent variable, time as the categorical variable and adjusted for Baseline WAL measurements, with compound symmetry covariance structure.
Time Frame: Baseline and Weeks 24 and 48
Population: TIO analysis set with available WAL measurements at Baseline and each time point.
Measure: Least Squares Mean (Standard Error); unit: arm lifts
Groups:
- Left Upper Extremity: Left arm lifts in participants who received burosumab at a starting dose of 0.3 mg/kg administered subcutaneously Q4W, titrated up to a maximum of 2.0 mg/kg Q2W.
- Right Upper Extremity: Right arm lifts in participants who received burosumab at a starting dose of 0.3 mg/kg administered subcutaneously Q4W, titrated up to a maximum of 2.0 mg/kg Q2W.
Arm/Group | Left Upper Extremity | Right Upper Extremity
Number analyzed (Participants) | 8 | 9
arm lifts
  Week 24 | -0.5 (1.09) | 0.6 (0.89)
  Week 48 | 0.1 (1.25) | 1.7 (1.17)
Statistical Analysis 1: Comparison: Left Upper Extremity; Week 24; Test type: Other; p = 0.6475, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 2: Comparison: Right Upper Extremity; Week 24; Test type: Other; p = 0.5319, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 3: Comparison: Left Upper Extremity; Week 48; Test type: Other; p = 0.9206, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 4: Comparison: Right Upper Extremity; Week 48; Test type: Other; p = 0.1530, GEE model; [statistical method as in outcome 28, analysis 1]

32. Secondary Outcome: Change From Baseline Over Time in Six-Minute Walk Test (6MWT)
Description: The 6MWT is a commonly used measure of mobility and was conducted in accordance with general principles set forth in the American Thoracic Society guidelines (ATS 2002). Participants were instructed to walk the length of a pre-measured course for 6 consecutive minutes (assistive devices could be used). The total distance walked at the end of 6 minutes was recorded in meters.
  Least squares means and standard errors were estimated from a generalized estimation equation (GEE) model which includes the change from Baseline as the dependent variable, time as the categorical variable and adjusted for Baseline 6MWT measurement, with compound symmetry covariance structure.
Time Frame: Baseline and Weeks 24 and 48
Population: TIO analysis set with available 6MWT measurements at Baseline and each time point. Six participants did not perform the test at Baseline as it was not included in the original protocol, and 2 participants were unable to perform the test due to underlying medical issues.
Measure: Least Squares Mean (Standard Error); unit: meters
Arm/Group | Burosumab
Number analyzed (Participants) | 6
meters
  Week 24 | 19.5 (15.64)
  Week 48 | 25.5 (16.58)
Statistical Analysis 1: Comparison: Burosumab; Week 24; Test type: Other; p = 0.2125, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 2: Comparison: Burosumab; Week 48; Test type: Other; p = 0.1241, GEE model; [statistical method as in outcome 28, analysis 1]

33. Secondary Outcome: Change From Baseline Over Time in Brief Pain Inventory (BPI) Worst Pain Score
Description: The Brief Pain Inventory (BPI) is a self-reported, pain-specific questionnaire with a recall period of 24 hours. Worst pain is defined as the answer to Question 3, in which participants rated their pain at its worst in the last 24 hours on a scale from 0 (no pain) to 10 (pain as bad as you can imagine).
  A negative change from Baseline score indicates improvement.
  Least squares means and standard errors were estimated from a generalized estimation equation (GEE) model which includes the change from Baseline as the dependent variable, time as the categorical variable and adjusted for Baseline BPI measurement, with compound symmetry covariance structure.
Time Frame: Baseline and Weeks 24, 48, 96, 144, 168, 192, 216, and 240
Population: TIO analysis set participants with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Burosumab
Number analyzed (Participants) | 14
score on a scale
  Week 24 | -0.6 (0.7)
  Week 48: number analyzed (Participants) | 13
  Week 48 | -0.9 (0.7)
  Week 96: number analyzed (Participants) | 12
  Week 96 | -0.7 (0.4)
  Week 144: number analyzed (Participants) | 11
  Week 144 | -1.1 (0.6)
  Week 168: number analyzed (Participants) | 10
  Week 168 | -0.9 (0.7)
  Week 192: number analyzed (Participants) | 10
  Week 192 | -0.9 (0.6)
  Week 216: number analyzed (Participants) | 7
  Week 216 | -0.9 (0.8)
  Week 240: number analyzed (Participants) | 7
  Week 240 | -0.9 (0.9)
Statistical Analysis 1: Comparison: Burosumab; Week 24; Test type: Other; p = 0.410, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 2: Comparison: Burosumab; Week 48; Test type: Other; p = 0.210, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 3: Comparison: Burosumab; Week 96; Test type: Other; p = 0.060, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 4: Comparison: Burosumab; Week 144; Test type: Other; p = 0.076, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 5: Comparison: Burosumab; Week 168; Test type: Other; p = 0.171, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 6: Comparison: Burosumab; Week 192; Test type: Other; p = 0.141, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 7: Comparison: Burosumab; Week 216; Test type: Other; p = 0.263, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 8: Comparison: Burosumab; Week 240; Test type: Other; p = 0.320, GEE model; [statistical method as in outcome 28, analysis 1]

34. Secondary Outcome: Change From Baseline Over Time in Brief Pain Inventory (BPI) Pain Severity Score
Description: The Brief Pain Inventory (BPI) is a self-reported, pain-specific questionnaire with a recall period of 24 hours.
  Pain severity is defined as the average of 4 questions (Questions 3 through 6) assessing worst pain, least pain, average pain, and pain right now, rated on a scale from 0 (no pain) to 10 (pain as bad as you can imagine). Mild pain is defined as a score of 1 to 4, moderate pain is defined as a score of 5 to 6, and severe pain is defined as a score of 7 to 10. A negative change from Baseline score indicates improvement.
  Least squares means and standard errors were estimated from a generalized estimation equation (GEE) model which includes the change from Baseline as the dependent variable, time as the categorical variable and adjusted for Baseline BPI measurement, with compound symmetry covariance structure.
Time Frame: Baseline and Weeks 24, 48, 96, 144, 168, 192, 216, and 240
Population: TIO analysis set participants with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Burosumab
Number analyzed (Participants) | 14
score on a scale
  Week 24 | -0.51 (0.62)
  Week 48: number analyzed (Participants) | 13
  Week 48 | -0.87 (0.66)
  Week 96: number analyzed (Participants) | 12
  Week 96 | -0.62 (0.38)
  Week 144: number analyzed (Participants) | 11
  Week 144 | -0.99 (0.42)
  Week 168: number analyzed (Participants) | 10
  Week 168 | -1.21 (0.40)
  Week 192: number analyzed (Participants) | 10
  Week 192 | -0.81 (0.66)
  Week 216: number analyzed (Participants) | 7
  Week 216 | -0.75 (0.63)
  Week 240: number analyzed (Participants) | 7
  Week 240 | -0.91 (0.76)
Statistical Analysis 1: Comparison: Burosumab; Week 24; Test type: Other; p = 0.407, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 2: Comparison: Burosumab; Week 48; Test type: Other; p = 0.192, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 3: Comparison: Burosumab; Week 96; Test type: Other; p = 0.106, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 4: Comparison: Burosumab; Week 144; Test type: Other; p = 0.020, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 5: Comparison: Burosumab; Week 168; Test type: Other; p = 0.002, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 6: Comparison: Burosumab; Week 192; Test type: Other; p = 0.220, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 7: Comparison: Burosumab; Week 216; Test type: Other; p = 0.230, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 8: Comparison: Burosumab; Week 240; Test type: Other; p = 0.232, GEE model; [statistical method as in outcome 28, analysis 1]

35. Secondary Outcome: Change From Baseline Over Time in Brief Pain Inventory (BPI) Pain Interference Score
Description: The Brief Pain Inventory (BPI) is a self-reported, pain-specific questionnaire with a recall period of 24 hours.
  Pain interference is defined as the average of 7 questions (9A through 9G) regarding the extent to which pain interfered with daily activities, including general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life in the last 24 hours, rated on a scale from 0 (does not interfere) to 10 (completely interferes).
  A negative change from Baseline score indicates improvement. Least squares means and standard errors were estimated from a generalized estimation equation (GEE) model which includes the change from Baseline as the dependent variable, time as the categorical variable and adjusted for Baseline BPI measurement, with compound symmetry covariance structure.
Time Frame: Baseline and Weeks 24, 48, 96, 144, 168, 192, 216, and 240
Population: TIO analysis set participants with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Burosumab
Number analyzed (Participants) | 14
score on a scale
  Week 24 | -1.15 (0.66)
  Week 48: number analyzed (Participants) | 13
  Week 48 | -1.09 (0.80)
  Week 96: number analyzed (Participants) | 12
  Week 96 | -1.08 (0.55)
  Week 144: number analyzed (Participants) | 11
  Week 144 | -1.46 (0.61)
  Week 168: number analyzed (Participants) | 10
  Week 168 | -1.76 (0.37)
  Week 192: number analyzed (Participants) | 10
  Week 192 | -1.11 (0.58)
  Week 216: number analyzed (Participants) | 7
  Week 216 | -1.56 (0.87)
  Week 240: number analyzed (Participants) | 7
  Week 240 | -2.00 (1.10)
Statistical Analysis 1: Comparison: Burosumab; Week 24; Test type: Other; p = 0.082, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 2: Comparison: Burosumab; Week 48; Test type: Other; p = 0.176, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 3: Comparison: Burosumab; Week 96; Test type: Other; p = 0.047, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 4: Comparison: Burosumab; Week 144; Test type: Other; p = 0.017, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 5: Comparison: Burosumab; Week 168; Test type: Other; p = 0.000, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 6: Comparison: Burosumab; Week 192; Test type: Other; p = 0.057, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 7: Comparison: Burosumab; Week 216; Test type: Other; p = 0.071, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 8: Comparison: Burosumab; Week 240; Test type: Other; p = 0.070, GEE model; [statistical method as in outcome 28, analysis 1]

36. Secondary Outcome: Change From Baseline Over Time in Brief Fatigue Inventory (BFI) Worst Fatigue Score
Description: The Brief Fatigue Inventory (BFI) is a self-reported questionnaire consisting of 9 items related to fatigue that are rated on a 0 to 10 numerical rating scale with a recall period of 24 hours.
  Worst fatigue is defined as the answer to Question 3 in which participants rated their fatigue at its worst in the last 24 hours on a scale from 0 (no fatigue) to 10 (as bad as you can imagine).
  A negative change from Baseline score indicates improvement. Least squares means and standard errors were estimated from a generalized estimation equation (GEE) model which includes the change from Baseline as the dependent variable, time as the categorical variable and adjusted for Baseline BFI measurement, with compound symmetry covariance structure.
Time Frame: Baseline and Weeks 24, 48, 96, 144, 168, 192, 216, and 240
Population: TIO analysis set participants with available data at Baseline and each time point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Burosumab
Number analyzed (Participants) | 13
score on a scale
  Week 24 | -1.3 (0.5)
  Week 48: number analyzed (Participants) | 12
  Week 48 | -0.9 (0.8)
  Week 96: number analyzed (Participants) | 11
  Week 96 | -1.0 (0.5)
  Week 144: number analyzed (Participants) | 10
  Week 144 | -0.9 (0.6)
  Week 168: number analyzed (Participants) | 9
  Week 168 | -1.6 (0.6)
  Week 192: number analyzed (Participants) | 9
  Week 192 | -1.0 (0.4)
  Week 216: number analyzed (Participants) | 6
  Week 216 | -2.1 (0.9)
  Week 240: number analyzed (Participants) | 6
  Week 240 | -2.6 (0.9)
Statistical Analysis 1: Comparison: Burosumab; Week 24; Test type: Other; p = 0.014, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 2: Comparison: Burosumab; Week 48; Test type: Other; p = 0.309, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 3: Comparison: Burosumab; Week 96; Test type: Other; p = 0.036, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 4: Comparison: Burosumab; Week 144; Test type: Other; p = 0.096, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 5: Comparison: Burosumab; Week 168; Test type: Other; p = 0.005, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 6: Comparison: Burosumab; Week 192; Test type: Other; p = 0.022, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 7: Comparison: Burosumab; Week 216; Test type: Other; p = 0.022, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 8: Comparison: Burosumab; Week 240; Test type: Other; p = 0.004, GEE model; [statistical method as in outcome 28, analysis 1]

37. Secondary Outcome: Change From Baseline Over Time in Brief Fatigue Inventory (BFI) Fatigue Severity Score
Description: The Brief Fatigue Inventory (BFI) is a self-reported questionnaire consisting of 9 items related to fatigue that are rated on a 0 to 10 numerical rating scale with a recall period of 24 hours.
  Fatigue severity is defined as the average of 3 questions (Questions 1 through 3) assessing fatigue right now, usual level of fatigue, and worst fatigue, rated on a scale from 0 (no fatigue) to 10 (as bad as you can imagine).
  A negative change from Baseline score indicates improvement.
  Least squares means and standard errors were estimated from a generalized estimation equation (GEE) model which includes the change from Baseline as the dependent variable, time as the categorical variable and adjusted for Baseline BFI measurement, with compound symmetry covariance structure.
Time Frame: Baseline and Weeks 24, 48, 96, 144, 168, 192, 216, and 240
Population: TIO analysis set participants with available data at Baseline and each time point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Burosumab
Number analyzed (Participants) | 13
score on a scale
  Week 24 | -1.47 (0.53)
  Week 48: number analyzed (Participants) | 12
  Week 48 | -1.31 (0.56)
  Week 96: number analyzed (Participants) | 11
  Week 96 | -1.58 (0.43)
  Week 144: number analyzed (Participants) | 10
  Week 144 | -1.44 (0.53)
  Week 168: number analyzed (Participants) | 9
  Week 168 | -2.34 (0.43)
  Week 192: number analyzed (Participants) | 9
  Week 192 | -1.62 (0.43)
  Week 216: number analyzed (Participants) | 6
  Week 216 | -2.62 (0.85)
  Week 240: number analyzed (Participants) | 6
  Week 240 | -2.57 (0.81)
Statistical Analysis 1: Comparison: Burosumab; Week 24; Test type: Other; p = 0.005, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 2: Comparison: Burosumab; Week 48; Test type: Other; p = 0.019, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 3: Comparison: Burosumab; Week 96; Test type: Other; p < 0.001, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 4: Comparison: Burosumab; Week 144; Test type: Other; p = 0.006, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 5: Comparison: Burosumab; Week 168; Test type: Other; p < 0.001, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 6: Comparison: Burosumab; Week 192; Test type: Other; p < 0.001, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 7: Comparison: Burosumab; Week 216; Test type: Other; p = 0.002, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 8: Comparison: Burosumab; Week 240; Test type: Other; p = 0.002, GEE model; [statistical method as in outcome 28, analysis 1]

38. Secondary Outcome: Change From Baseline Over Time in Brief Fatigue Inventory (BFI) Fatigue Interference Score
Description: The Brief Fatigue Inventory (BFI) is a self-reported questionnaire consisting of 9 items related to fatigue that are rated on a 0 to 10 numerical rating scale with a recall period of 24 hours.
  The fatigue interference score is defined as the average of 6 questions (Questions 4A through 4F) regarding the extent to which fatigue interfered with daily activities, including general activity, mood, walking ability, work, relations with others, and enjoyment of life in the last 24 hours, rated on a scale from 0 (does not interfere) to 10 (completely interferes).
  A negative change from Baseline score indicates improvement. Least squares means and standard errors were estimated from a generalized estimation equation (GEE) model which includes the change from Baseline as the dependent variable, time as the categorical variable and adjusted for Baseline BFI measurement, with compound symmetry covariance structure.
Time Frame: Baseline and Weeks 24, 48, 96, 144, 168, 192, 216, and 240
Population: TIO analysis set participants with available data at Baseline and each time point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Burosumab
Number analyzed (Participants) | 13
score on a scale
  Week 24 | -1.57 (0.65)
  Week 48: number analyzed (Participants) | 12
  Week 48 | -1.88 (0.66)
  Week 96: number analyzed (Participants) | 11
  Week 96 | -1.98 (0.47)
  Week 144: number analyzed (Participants) | 10
  Week 144 | -1.67 (0.44)
  Week 168: number analyzed (Participants) | 9
  Week 168 | -2.20 (0.38)
  Week 192: number analyzed (Participants) | 9
  Week 192 | -1.24 (0.59)
  Week 216: number analyzed (Participants) | 6
  Week 216 | -2.72 (1.02)
  Week 240: number analyzed (Participants) | 6
  Week 240 | -3.00 (1.14)
Statistical Analysis 1: Comparison: Burosumab; Week 24; Test type: Other; p = 0.016, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 2: Comparison: Burosumab; Week 48; Test type: Other; p = 0.004, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 3: Comparison: Burosumab; Week 96; Test type: Other; p < 0.001, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 4: Comparison: Burosumab; Week 144; Test type: Other; p < 0.001, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 5: Comparison: Burosumab; Week 168; Test type: Other; p < 0.001, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 6: Comparison: Burosumab; Week 192; Test type: Other; p = 0.036, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 7: Comparison: Burosumab; Week 216; Test type: Other; p = 0.008, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 8: Comparison: Burosumab; Week 240; Test type: Other; p = 0.008, GEE model; [statistical method as in outcome 28, analysis 1]

39. Secondary Outcome: Change From Baseline Over Time in Brief Fatigue Inventory (BFI) Global Fatigue Score
Description: The Brief Fatigue Inventory (BFI) is a self-reported questionnaire consisting of 9 items related to fatigue that are rated on a 0 to 10 numerical rating scale with a recall period of 24 hours. The first 3 questions measure fatigue severity and the next 6 questions assess the impact of fatigue on daily activities.
  The global fatigue score is defined as the average of all 9 questions on the BFI including severity and interference, and ranges from from 0 to 10, where higher scores correspond to greater levels of fatigue.
  A negative change from Baseline score indicates improvement. Least squares means and standard errors were estimated from a generalized estimation equation (GEE) model which includes the change from Baseline as the dependent variable, time as the categorical variable and adjusted for Baseline BFI measurement, with compound symmetry covariance structure.
Time Frame: Baseline and Weeks 24, 48, 96, 144, 168, 192, 216, and 240
Population: TIO analysis set participants with available data at Baseline and each time point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Burosumab
Number analyzed (Participants) | 13
score on a scale
  Week 24 | -1.54 (0.56)
  Week 48: number analyzed (Participants) | 12
  Week 48 | -1.66 (0.56)
  Week 96: number analyzed (Participants) | 11
  Week 96 | -1.83 (0.44)
  Week 144: number analyzed (Participants) | 10
  Week 144 | -1.58 (0.44)
  Week 168: number analyzed (Participants) | 9
  Week 168 | -2.23 (0.37)
  Week 192: number analyzed (Participants) | 9
  Week 192 | -1.34 (0.50)
  Week 216: number analyzed (Participants) | 6
  Week 216 | -2.66 (0.95)
  Week 240: number analyzed (Participants) | 6
  Week 240 | -2.83 (1.02)
Statistical Analysis 1: Comparison: Burosumab; Week 24; Test type: Other; p = 0.006, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 2: Comparison: Burosumab; Week 48; Test type: Other; p = 0.003, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 3: Comparison: Burosumab; Week 96; Test type: Other; p < 0.001, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 4: Comparison: Burosumab; Week 144; Test type: Other; p < 0.001, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 5: Comparison: Burosumab; Week 168; Test type: Other; p < 0.001, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 6: Comparison: Burosumab; Week 192; Test type: Superiority; p = 0.007, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 7: Comparison: Burosumab; Week 216; Test type: Other; p = 0.005, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 8: Comparison: Burosumab; Week 240; Test type: Other; p = 0.006, GEE model; [statistical method as in outcome 28, analysis 1]

40. Secondary Outcome: Change From Baseline Over Time in 36-Item Short Form Health Survey (SF-36) Physical Component Summary Score
Description: The SF-36 v2 is a self-administered questionnaire that measures the impact of disease on overall quality of life during the past 4 weeks. The SF-36 consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health).
  The physical component summary score (PCS) is a weighted combination of the 8 subscales with positive weighting for physical functioning, role-physical, bodily pain, and general health. The PCS was calculated using norm-based scoring so that 50 is the average score and the standard deviation equals 10. Higher scores are associated with better functioning/quality of life; a positive change from Baseline score indicates an improvement.
  LS means and SEs were estimated from a GEE model which includes the change from Baseline as the dependent variable, time as the categorical variable and adjusted for Baseline SF-36, with compound symmetry covariance struct
Time Frame: Baseline and Weeks 24, 48, 96, 144, 168, 192, 216, and 240
Population: TIO analysis set participants with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Burosumab
Number analyzed (Participants) | 14
score on a scale
  Week 24 | 3.71 (1.42)
  Week 48: number analyzed (Participants) | 13
  Week 48 | 5.43 (2.33)
  Week 96: number analyzed (Participants) | 12
  Week 96 | 2.75 (1.37)
  Week 144: number analyzed (Participants) | 10
  Week 144 | 7.98 (2.40)
  Week 168: number analyzed (Participants) | 10
  Week 168 | 5.20 (2.14)
  Week 192: number analyzed (Participants) | 10
  Week 192 | 3.82 (2.49)
  Week 216: number analyzed (Participants) | 7
  Week 216 | 6.17 (2.17)
  Week 240: number analyzed (Participants) | 7
  Week 240 | 5.82 (2.45)
Statistical Analysis 1: Comparison: Burosumab; Week 24; Test type: Other; p = 0.009, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 2: Comparison: Burosumab; Week 48; Test type: Other; p = 0.020, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 3: Comparison: Burosumab; Week 96; Test type: Other; p = 0.044, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 4: Comparison: Burosumab; Week 144; Test type: Other; p < 0.001, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 5: Comparison: Burosumab; Week 168; Test type: Other; p = 0.015, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 6: Comparison: Burosumab; Week 192; Test type: Other; p = 0.125, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 7: Comparison: Burosumab; Week 216; Test type: Other; p = 0.004, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 8: Comparison: Burosumab; Week 240; Test type: Other; p = 0.018, GEE model; [statistical method as in outcome 28, analysis 1]

41. Secondary Outcome: Change From Baseline Over Time in 36-Item Short Form Health Survey (SF-36) Physical Functioning Domain Score
Description: The SF-36 v2 is a self-administered questionnaire that measures the impact of disease on overall quality of life during the past 4 weeks. The SF-36 consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health).
  The physical functioning (PF) domain includes 10 questions that assess limitations in physical activities because of health problems. The PF domain score was calculated using norm-based scoring so that 50 is the average score and the standard deviation equals 10. Higher scores are associated with better functioning/quality of life; a positive change from Baseline score indicates an improvement.
  LS means and SEs were estimated from a GEE model which includes the change from Baseline as the dependent variable, time as the categorical variable and adjusted for Baseline SF-36, with compound symmetry covariance structure.
Time Frame: Baseline and Weeks 24, 48, 96, 144, 168, 192, 216, and 240
Population: TIO analysis set participants with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Burosumab
Number analyzed (Participants) | 14
score on a scale
  Week 24 | 2.29 (1.58)
  Week 48: number analyzed (Participants) | 13
  Week 48 | 2.63 (2.51)
  Week 96: number analyzed (Participants) | 12
  Week 96 | 3.77 (1.58)
  Week 144: number analyzed (Participants) | 11
  Week 144 | 7.89 (2.00)
  Week 168: number analyzed (Participants) | 10
  Week 168 | 5.50 (2.24)
  Week 192: number analyzed (Participants) | 10
  Week 192 | 3.02 (2.04)
  Week 216: number analyzed (Participants) | 7
  Week 216 | 6.75 (1.96)
  Week 240: number analyzed (Participants) | 7
  Week 240 | 4.56 (3.11)
Statistical Analysis 1: Comparison: Burosumab; Week 24; Test type: Other; p = 0.148, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 2: Comparison: Burosumab; Week 48; Test type: Other; p = 0.295, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 3: Comparison: Burosumab; Week 96; Test type: Other; p = 0.005, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 4: Comparison: Burosumab; Week 144; Test type: Other; p < 0.001, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 5: Comparison: Burosumab; Week 168; Test type: Other; p = 0.014, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 6: Comparison: Burosumab; Week 192; Test type: Other; p = 0.140, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 7: Comparison: Burosumab; Week 216; Test type: Other; p < 0.001, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 8: Comparison: Burosumab; Week 240; Test type: Other; p = 0.142, GEE model; [statistical method as in outcome 28, analysis 1]

42. Secondary Outcome: Change From Baseline Over Time in 36-Item Short Form Health Survey (SF-36) Role Physical Domain Score
Description: The SF-36 v2 is a self-administered questionnaire that measures the impact of disease on overall quality of life during the past 4 weeks. The SF-36 consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health).
  The role-physical (RP) domain includes 4 questions that assess limitations in usual role activities because of physical health problems. The RP domain score was calculated using norm-based scoring so that 50 is the average score and the standard deviation equals 10. Higher scores are associated with better functioning/quality of life; a positive change from Baseline score indicates an improvement.
  LS means and SEs were estimated from a GEE model which includes the change from Baseline as the dependent variable, time as the categorical variable and adjusted for Baseline SF-36, with compound symmetry covariance structure.
Time Frame: Baseline and Weeks 24, 48, 96, 144, 168, 192, 216, and 240
Population: TIO analysis set participants with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Burosumab
Number analyzed (Participants) | 14
score on a scale
  Week 24 | 4.85 (1.74)
  Week 48: number analyzed (Participants) | 13
  Week 48 | 5.00 (2.83)
  Week 96: number analyzed (Participants) | 12
  Week 96 | 3.25 (1.63)
  Week 144: number analyzed (Participants) | 10
  Week 144 | 5.53 (2.81)
  Week 168: number analyzed (Participants) | 10
  Week 168 | 5.70 (1.93)
  Week 192: number analyzed (Participants) | 10
  Week 192 | 5.03 (2.80)
  Week 216: number analyzed (Participants) | 7
  Week 216 | 4.82 (3.01)
  Week 240: number analyzed (Participants) | 7
  Week 240 | 8.99 (3.28)
Statistical Analysis 1: Comparison: Burosumab; Week 24; Test type: Other; p = 0.005, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 2: Comparison: Burosumab; Week 48; Test type: Other; p = 0.077, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 3: Comparison: Burosumab; Week 96; Test type: Other; p = 0.046, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 4: Comparison: Burosumab; Week 144; Test type: Other; p = 0.049, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 5: Comparison: Burosumab; Week 168; Test type: Other; p = 0.003, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 6: Comparison: Burosumab; Week 192; Test type: Other; p = 0.073, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 7: Comparison: Burosumab; Week 216; Test type: Other; p = 0.109, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 8: Comparison: Burosumab; Week 240; Test type: Other; p = 0.006, GEE model; [statistical method as in outcome 28, analysis 1]

43. Secondary Outcome: Change From Baseline Over Time in 36-Item Short Form Health Survey (SF-36) Bodily Pain Domain Score
Description: The SF-36 v2 is a self-administered questionnaire that measures the impact of disease on overall quality of life during the past 4 weeks. The SF-36 consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health).
  The bodily pain (BP) domain includes 2 questions that assess pain level and impact of pain on normal work. The BP domain score was calculated using norm-based scoring so that 50 is the average score and the standard deviation equals 10. Higher scores are associated with better functioning/quality of life; a positive change from Baseline score indicates an improvement.
  LS means and SEs were estimated from a GEE model which includes the change from Baseline as the dependent variable, time as the categorical variable and adjusted for Baseline SF-36, with compound symmetry covariance structure.
Time Frame: Baseline and Weeks 24, 48, 96, 144, 168, 192, 216, and 240
Population: TIO analysis set participants with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Burosumab
Number analyzed (Participants) | 14
score on a scale
  Week 24 | 1.61 (1.65)
  Week 48: number analyzed (Participants) | 13
  Week 48 | 3.61 (1.48)
  Week 96: number analyzed (Participants) | 12
  Week 96 | 2.52 (1.08)
  Week 144: number analyzed (Participants) | 11
  Week 144 | 5.40 (1.90)
  Week 168: number analyzed (Participants) | 10
  Week 168 | 5.01 (2.16)
  Week 192: number analyzed (Participants) | 10
  Week 192 | 4.92 (2.81)
  Week 216: number analyzed (Participants) | 7
  Week 216 | 6.64 (1.88)
  Week 240: number analyzed (Participants) | 7
  Week 240 | 6.59 (2.20)
Statistical Analysis 1: Comparison: Burosumab; Week 24; Test type: Other; p = 0.328, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 2: Comparison: Burosumab; Week 48; Test type: Other; p = 0.015, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 3: Comparison: Burosumab; Week 96; Test type: Other; p = 0.020, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 4: Comparison: Burosumab; Week 144; Test type: Other; p = 0.004, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 5: Comparison: Burosumab; Week 168; Test type: Other; p = 0.021, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 6: Comparison: Burosumab; Week 192; Test type: Other; p = 0.080, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 7: Comparison: Burosumab; Week 216; Test type: Other; p < 0.001, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 8: Comparison: Burosumab; Week 240; Test type: Other; p = 0.003, GEE model; [statistical method as in outcome 28, analysis 1]

44. Secondary Outcome: Change From Baseline Over Time in 36-Item Short Form Health Survey (SF-36) General Health Perceptions Domain Score
Description: The SF-36 v2 is a self-administered questionnaire that measures the impact of disease on overall quality of life during the past 4 weeks. The SF-36 consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health).
  The general health perceptions (GH) domain includes 5 questions that assess participants' perception of their own general health. The GH domain score was calculated using norm-based scoring so that 50 is the average score and the standard deviation equals 10. Higher scores are associated with better functioning/quality of life; a positive change from Baseline score indicates an improvement.
  LS means and SEs were estimated from a GEE model which includes the change from Baseline as the dependent variable, time as the categorical variable and adjusted for Baseline SF-36, with compound symmetry covariance structure.
Time Frame: Baseline and Weeks 24, 48, 96, 144, 168, 192, 216, and 240
Population: TIO analysis set participants with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Burosumab
Number analyzed (Participants) | 14
score on a scale
  Week 24 | 2.38 (1.88)
  Week 48: number analyzed (Participants) | 13
  Week 48 | 6.09 (2.28)
  Week 96: number analyzed (Participants) | 12
  Week 96 | 1.03 (1.96)
  Week 144: number analyzed (Participants) | 11
  Week 144 | 3.12 (2.64)
  Week 168: number analyzed (Participants) | 10
  Week 168 | -0.32 (2.51)
  Week 192: number analyzed (Participants) | 10
  Week 192 | -1.60 (2.94)
  Week 216: number analyzed (Participants) | 7
  Week 216 | -1.51 (2.05)
  Week 240: number analyzed (Participants) | 7
  Week 240 | 1.81 (3.30)
Statistical Analysis 1: Comparison: Burosumab; Week 24; Test type: Other; p = 0.207, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 2: Comparison: Burosumab; Week 48; Test type: Other; p = 0.008, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 3: Comparison: Burosumab; Week 96; Test type: Other; p = 0.598, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 4: Comparison: Burosumab; Week 144; Test type: Other; p = 0.237, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 5: Comparison: Burosumab; Week 168; Test type: Other; p = 0.899, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 6: Comparison: Burosumab; Week 192; Test type: Other; p = 0.585, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 7: Comparison: Burosumab; Week 216; Test type: Other; p = 0.461, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 8: Comparison: Burosumab; Week 240; Test type: Other; p = 0.583, GEE model; [statistical method as in outcome 28, analysis 1]

45. Secondary Outcome: Change From Baseline Over Time in 36-Item Short Form Health Survey (SF-36) Mental Component Summary Score
Description: The SF-36 v2 is a self-administered questionnaire that measures the impact of disease on overall quality of life during the past 4 weeks. The SF-36 consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health).
  The mental component summary score (MCS) is a weighted combination of the 8 subscales with positive weighting for vitality, social function, role limitations due to emotional problems, and mental health. The MCS was calculated using norm-based scoring so that 50 is the average score and the standard deviation equals 10. Higher scores are associated with better functioning/quality of life; a positive change from Baseline indicates an improvement.
  LS means and SEs were estimated from a GEE model which includes the change from Baseline as the dependent variable, time as the categorical variable and adjusted for Baseline SF-36, with compound symmetry covariance structure.
Time Frame: Baseline and Weeks 24, 48, 96, 144, 168, 192, 216, and 240
Population: TIO analysis set participants with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Burosumab
Number analyzed (Participants) | 14
score on a scale
  Week 24 | 1.07 (2.38)
  Week 48: number analyzed (Participants) | 13
  Week 48 | 1.37 (2.47)
  Week 96: number analyzed (Participants) | 12
  Week 96 | 3.91 (2.53)
  Week 144: number analyzed (Participants) | 10
  Week 144 | -0.85 (2.29)
  Week 168: number analyzed (Participants) | 10
  Week 168 | 2.05 (1.81)
  Week 192: number analyzed (Participants) | 10
  Week 192 | 0.55 (2.95)
  Week 216: number analyzed (Participants) | 7
  Week 216 | 0.51 (2.67)
  Week 240: number analyzed (Participants) | 7
  Week 240 | 5.13 (3.59)
Statistical Analysis 1: Comparison: Burosumab; Week 24; Test type: Other; p = 0.654, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 2: Comparison: Burosumab; Week 48; Test type: Other; p = 0.579, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 3: Comparison: Burosumab; Week 96; Test type: Other; p = 0.123, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 4: Comparison: Burosumab; Week 144; Test type: Other; p = 0.712, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 5: Comparison: Burosumab; Week 168; Test type: Other; p = 0.258, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 6: Comparison: Burosumab; Week 192; Test type: Other; p = 0.851, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 7: Comparison: Burosumab; Week 216; Test type: Other; p = 0.849, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 8: Comparison: Burosumab; Week 240; Test type: Other; p = 0.153, GEE model; [statistical method as in outcome 28, analysis 1]

46. Secondary Outcome: Change From Baseline Over Time in 36-Item Short Form Health Survey (SF-36) Vitality Domain Score
Description: The SF-36 v2 is a self-administered questionnaire that measures the impact of disease on overall quality of life during the past 4 weeks. The SF-36 consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health).
  The vitality (VT) domain includes 4 questions that assess energy levels and fatigue. The VT domain score was calculated using norm-based scoring so that 50 is the average score and the standard deviation equals 10. Higher scores are associated with better functioning/quality of life; a positive change from Baseline score indicates an improvement.
  LS means and SEs were estimated from a GEE model which includes the change from Baseline as the dependent variable, time as the categorical variable and adjusted for Baseline SF-36, with compound symmetry covariance structure.
Time Frame: Baseline and Weeks 24, 48, 96, 144, 168, 192, 216, and 240
Population: TIO analysis set participants with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Burosumab
Number analyzed (Participants) | 14
score on a scale
  Week 24 | 5.98 (1.96)
  Week 48: number analyzed (Participants) | 13
  Week 48 | 5.27 (2.42)
  Week 96: number analyzed (Participants) | 12
  Week 96 | 6.71 (2.64)
  Week 144: number analyzed (Participants) | 11
  Week 144 | 3.05 (2.30)
  Week 168: number analyzed (Participants) | 10
  Week 168 | 6.04 (2.74)
  Week 192: number analyzed (Participants) | 10
  Week 192 | 2.78 (2.85)
  Week 216: number analyzed (Participants) | 7
  Week 216 | 6.79 (3.77)
  Week 240: number analyzed (Participants) | 7
  Week 240 | 8.06 (4.03)
Statistical Analysis 1: Comparison: Burosumab; Week 24; Test type: Other; p = 0.002, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 2: Comparison: Burosumab; Week 48; Test type: Other; p = 0.030, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 3: Comparison: Burosumab; Week 96; Test type: Other; p = 0.011, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 4: Comparison: Burosumab; Week 144; Test type: Other; p = 0.186, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 5: Comparison: Burosumab; Week 168; Test type: Other; p = 0.027, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 6: Comparison: Burosumab; Week 192; Test type: Other; p = 0.330, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 7: Comparison: Burosumab; Week 216; Test type: Other; p = 0.072, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 8: Comparison: Burosumab; Week 240; Test type: Other; p = 0.045, GEE model; [statistical method as in outcome 28, analysis 1]

47. Secondary Outcome: Change From Baseline Over Time in 36-Item Short Form Health Survey (SF-36) Social Functioning Domain Score
Description: The SF-36 v2 is a self-administered questionnaire that measures the impact of disease on overall quality of life during the past 4 weeks. The SF-36 consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health).
  The social functioning (SF) domain includes 2 questions that assess limitations in social activities because of physical health or emotional problems. The SF domain score was calculated using norm-based scoring so that 50 is the average score and the standard deviation equals 10. Higher scores are associated with better functioning/quality of life; a positive change from Baseline score indicates an improvement.
  LS means and SEs were estimated from a GEE model which includes the change from Baseline as the dependent variable, time as the categorical variable and adjusted for Baseline SF-36, with compound symmetry covariance structure.
Time Frame: Baseline and Weeks 24, 48, 96, 144, 168, 192, 216, and 240
Population: TIO analysis set participants with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Burosumab
Number analyzed (Participants) | 14
score on a scale
  Week 24 | 2.02 (2.24)
  Week 48: number analyzed (Participants) | 13
  Week 48 | 5.54 (2.48)
  Week 96: number analyzed (Participants) | 12
  Week 96 | 4.63 (1.34)
  Week 144: number analyzed (Participants) | 11
  Week 144 | 3.22 (2.71)
  Week 168: number analyzed (Participants) | 10
  Week 168 | 5.34 (2.06)
  Week 192: number analyzed (Participants) | 10
  Week 192 | 2.84 (2.62)
  Week 216: number analyzed (Participants) | 7
  Week 216 | 4.15 (2.08)
  Week 240: number analyzed (Participants) | 7
  Week 240 | 6.30 (2.98)
Statistical Analysis 1: Comparison: Burosumab; Week 24; Test type: Other; p = 0.369, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 2: Comparison: Burosumab; Week 48; Test type: Other; p = 0.026, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 3: Comparison: Burosumab; Week 96; Test type: Other; p < 0.001, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 4: Comparison: Burosumab; Week 144; Test type: Other; p = 0.235, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 5: Comparison: Burosumab; Week 168; Test type: Other; p = 0.009, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 6: Comparison: Burosumab; Week 192; Test type: Other; p = 0.278, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 7: Comparison: Burosumab; Week 216; Test type: Other; p = 0.046, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 8: Comparison: Burosumab; Week 240; Test type: Other; p = 0.035, GEE model; [statistical method as in outcome 28, analysis 1]

48. Secondary Outcome: Change From Baseline Over Time in 36-Item Short Form Health Survey (SF-36) Role Emotional Domain Score
Description: The SF-36 v2 is a self-administered questionnaire that measures the impact of disease on overall quality of life during the past 4 weeks. The SF-36 consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health).
  The role-emotional (RE) domain includes 3 questions that assess limitations in usual role activities because of emotional problems. The RE domain score was calculated using norm-based scoring so that 50 is the average score and the standard deviation equals 10. Higher scores are associated with better functioning/quality of life; a positive change from Baseline score indicates an improvement.
  LS means and SEs were estimated from a GEE model which includes the change from Baseline as the dependent variable, time as the categorical variable and adjusted for Baseline SF-36, with compound symmetry covariance structure.
Time Frame: Baseline and Weeks 24, 48, 96, 144, 168, 192, 216, and 240
Population: TIO analysis set participants with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Burosumab
Number analyzed (Participants) | 14
score on a scale
  Week 24 | 1.52 (1.98)
  Week 48: number analyzed (Participants) | 13
  Week 48 | 1.13 (2.72)
  Week 96: number analyzed (Participants) | 12
  Week 96 | 6.73 (3.03)
  Week 144: number analyzed (Participants) | 10
  Week 144 | 2.10 (2.60)
  Week 168: number analyzed (Participants) | 10
  Week 168 | 4.90 (2.22)
  Week 192: number analyzed (Participants) | 10
  Week 192 | 3.51 (3.47)
  Week 216: number analyzed (Participants) | 7
  Week 216 | 3.56 (3.08)
  Week 240: number analyzed (Participants) | 7
  Week 240 | 6.04 (3.69)
Statistical Analysis 1: Comparison: Burosumab; Week 24; Test type: Other; p = 0.442, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 2: Comparison: Burosumab; Week 48; Test type: Other; p = 0.677, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 3: Comparison: Burosumab; Week 96; Test type: Other; p = 0.027, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 4: Comparison: Burosumab; Week 144; Test type: Other; p = 0.420, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 5: Comparison: Burosumab; Week 168; Test type: Superiority; p = 0.027, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 6: Comparison: Burosumab; Week 192; Test type: Other; p = 0.312, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 7: Comparison: Burosumab; Week 216; Test type: Other; p = 0.249, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 8: Comparison: Burosumab; Week 240; Test type: Other; p = 0.102, GEE model; [statistical method as in outcome 28, analysis 1]

49. Secondary Outcome: Change From Baseline Over Time in 36-Item Short Form Health Survey (SF-36) Mental Health Domain Score
Description: The SF-36 v2 is a self-administered questionnaire that measures the impact of disease on overall quality of life during the past 4 weeks. The SF-36 consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health).
  The mental health (MH) domain includes 5 questions that assess general mental health (psychological distress and well-being). The MH domain score was calculated using norm-based scoring so that 50 is the average score and the standard deviation equals 10. Higher scores are associated with better functioning/quality of life; a positive change from Baseline score indicates an improvement.
  LS means and SEs were estimated from a GEE model which includes the change from Baseline as the dependent variable, time as the categorical variable and adjusted for Baseline SF-36, with compound symmetry covariance structure.
Time Frame: Baseline and Weeks 24, 48, 96, 144, 168, 192, 216, and 240
Population: TIO analysis set participants with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Burosumab
Number analyzed (Participants) | 14
score on a scale
  Week 24 | -0.46 (2.54)
  Week 48: number analyzed (Participants) | 13
  Week 48 | -0.32 (2.48)
  Week 96: number analyzed (Participants) | 12
  Week 96 | -0.58 (2.12)
  Week 144: number analyzed (Participants) | 11
  Week 144 | -0.17 (1.97)
  Week 168: number analyzed (Participants) | 10
  Week 168 | -0.97 (1.61)
  Week 192: number analyzed (Participants) | 10
  Week 192 | -1.24 (2.23)
  Week 216: number analyzed (Participants) | 7
  Week 216 | -2.11 (2.87)
  Week 240: number analyzed (Participants) | 7
  Week 240 | 3.50 (3.10)
Statistical Analysis 1: Comparison: Burosumab; Week 24; Test type: Other; p = 0.856, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 2: Comparison: Burosumab; Week 48; Test type: Other; p = 0.898, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 3: Comparison: Burosumab; Week 96; Test type: Other; p = 0.785, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 4: Comparison: Burosumab; Week 144; Test type: Other; p = 0.932, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 5: Comparison: Burosumab; Week 168; Test type: Other; p = 0.545, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 6: Comparison: Burosumab; Week 192; Test type: Other; p = 0.580, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 7: Comparison: Burosumab; Week 216; Test type: Other; p = 0.462, GEE model; [statistical method as in outcome 28, analysis 1]
Statistical Analysis 8: Comparison: Burosumab; Week 240; Test type: Other; p = 0.260, GEE model; [statistical method as in outcome 28, analysis 1]

50. Other Pre Specified Outcome: Number of Participants With Adverse Events (AEs), Treatment Emergent AEs (TEAEs), Serious TEAEs, and TEAEs Leading to Discontinuation
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug, whether or not considered drug related. A serious AE was defined as an AE that at any dose, in the view of either the Investigator or Sponsor, results in any of the following outcomes: death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant incapacity or disability, a congenital anomaly/birth defect, or other important medical events (according to the investigator). An AE was considered a TEAE if it occurred on or after the first dose and was not present prior to the first dose, or it was present prior to the first dose but increased in severity during the study. Events were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0: grade 1 (mild), grade 2 (moderate), grade 3 (severe), grade 4 (life-threatening), grade 5 (death).
Time Frame: From first dose of study drug up to database lock date (July 07, 2021); median duration of treatment in the TIO analysis set was 1594.0 (range: 168-2106) days.
Population: TIO analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Burosumab
Number analyzed (Participants) | 14
Participants
  Any adverse event | 14
  Serious adverse events (SAEs) | 8
  Related adverse events | 9
  Serious related adverse events | 0
  Grade 3 or 4 adverse event | 8
  TEAE leading to study discontinuation | 0
  TEAE leading to treatment discontinuation | 1
  TEAE leading to death | 2

51. Other Pre Specified Outcome: Number of Participants With Anti-burosumab Antibodies
Time Frame: as for outcome 50
Population: TIO analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Burosumab
Number analyzed (Participants) | 14
Participants
  Anti-burosumab binding antibodies | 2
  Anti-burosumab neutralizing antibodies | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to database lock date (July 07, 2021); median duration of treatment in the TIO analysis set was 1594.0 (range: 168-2106) days.
Groups:
- KRN23 TIO: Participants with TIO received burosumab at a starting dose of 0.3 mg/kg administered subcutaneously (SC) every 4 weeks (Q4W). Doses may have been titrated up to a maximum of 2.0 mg/kg every 2 weeks (Q2W) in order to achieve fasting peak serum phosphorus levels within the target range of 2.5 to 4.0 mg/dL.
- KRN23 XLH and ENS: Participants with XLH and ENS received burosumab at a starting dose of 0.3 mg/kg administered subcutaneously (SC) every 4 weeks (Q4W). Doses may have been titrated up to a maximum of 2.0 mg/kg every 2 weeks (Q2W) in order to achieve fasting peak serum phosphorus levels within the target range of 2.5 to 4.0 mg/dL.
Arm/Group | KRN23 TIO | KRN23 XLH and ENS
All-Cause Mortality (participants affected / at risk) | 2/14 | 0/3
Serious Adverse Events (participants affected / at risk) | 8/14 | 0/3
Other Adverse Events (participants affected / at risk) | 14/14 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | KRN23 TIO (N=14) | KRN23 XLH and ENS (N=3)
Cardiac Arrest (Cardiac disorders) | 2 | 0
Pulseless Electrical Activity (Cardiac disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Multi-Organ Failure (General disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Septic Shock (Infections and infestations) | 1 | 0
Sialoadenitis (Infections and infestations) | 1 | 0
Tooth Abscess (Infections and infestations) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Metastases To Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour Compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pickwickian Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | KRN23 TIO (N=14) | KRN23 XLH and ENS (N=3)
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 2 | 0
Eyelid Ptosis (Eye disorders) | 1 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 2 | 0
Abdominal Distension (Gastrointestinal disorders) | 2 | 0
Abdominal Hernia (Gastrointestinal disorders) | 1 | 0
Abdominal Mass (Gastrointestinal disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 3 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 2 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 4 | 0
Dental Caries (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0
Hypoaesthesia Oral (Gastrointestinal disorders) | 1 | 0
Large Intestine Polyp (Gastrointestinal disorders) | 1 | 0
Localised Intraabdominal Fluid Collection (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 1
Poor Dental Condition (Gastrointestinal disorders) | 1 | 0
Retching (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 5 | 1
Adverse Drug Reaction (General disorders) | 0 | 1
Application Site Rash (General disorders) | 1 | 0
Asthenia (General disorders) | 2 | 0
Calcinosis (General disorders) | 1 | 0
Chest Pain (General disorders) | 1 | 0
Chills (General disorders) | 2 | 0
Fatigue (General disorders) | 3 | 0
Gait Disturbance (General disorders) | 1 | 0
Generalised Oedema (General disorders) | 1 | 0
Influenza Like Illness (General disorders) | 0 | 1
Injection Site Bruising (General disorders) | 1 | 0
Injection Site Erythema (General disorders) | 0 | 1
Injection Site Pain (General disorders) | 1 | 0
Injection Site Reaction (General disorders) | 2 | 0
Injection Site Swelling (General disorders) | 1 | 0
Medical Device Site Reaction (General disorders) | 1 | 0
Nodule (General disorders) | 1 | 0
Oedema Peripheral (General disorders) | 3 | 0
Pain (General disorders) | 4 | 1
Peripheral Swelling (General disorders) | 1 | 1
Pyrexia (General disorders) | 2 | 0
Ulcer (General disorders) | 0 | 1
Bile Duct Stone (Hepatobiliary disorders) | 1 | 0
Hepatic Cyst (Hepatobiliary disorders) | 1 | 0
Hepatic Lesion (Hepatobiliary disorders) | 1 | 0
Seasonal Allergy (Immune system disorders) | 1 | 1
Bronchitis (Infections and infestations) | 3 | 0
Conjunctivitis (Infections and infestations) | 1 | 0
Corona Virus Infection (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Gastrointestinal Infection (Infections and infestations) | 1 | 0
Gastrointestinal Viral Infection (Infections and infestations) | 1 | 0
Gingivitis (Infections and infestations) | 0 | 1
H1n1 Influenza (Infections and infestations) | 1 | 0
Incision Site Cellulitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 3 | 0
Nasopharyngitis (Infections and infestations) | 5 | 1
Oesophageal Candidiasis (Infections and infestations) | 1 | 0
Oral Candidiasis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1
Tooth Abscess (Infections and infestations) | 1 | 0
Tooth Infection (Infections and infestations) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 7 | 1
Urinary Tract Infection (Infections and infestations) | 4 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 | 1
Animal Bite (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 3 | 0
Fall (Injury, poisoning and procedural complications) | 4 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 0
Fibula Fracture (Injury, poisoning and procedural complications) | 1 | 0
Foot Fracture (Injury, poisoning and procedural complications) | 2 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0
Incision Site Rash (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Ligament Rupture (Injury, poisoning and procedural complications) | 1 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 3 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 1
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 1 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 3 | 1
Radiation Mucositis (Injury, poisoning and procedural complications) | 1 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 2 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 | 0
Scar (Injury, poisoning and procedural complications) | 1 | 0
Skin Abrasion (Injury, poisoning and procedural complications) | 1 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 0
Stress Fracture (Injury, poisoning and procedural complications) | 1 | 0
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 1
Tibia Fracture (Injury, poisoning and procedural complications) | 1 | 0
Tooth Fracture (Injury, poisoning and procedural complications) | 2 | 1
Tooth Injury (Injury, poisoning and procedural complications) | 1 | 0
Amylase Increased (Investigations) | 4 | 1
Blood Calcium Increased (Investigations) | 1 | 0
Blood Cholesterol Increased (Investigations) | 1 | 0
Blood Creatine Increased (Investigations) | 1 | 0
Blood Creatinine Increased (Investigations) | 1 | 0
Blood Glucose Increased (Investigations) | 1 | 0
Blood Parathyroid Hormone Increased (Investigations) | 1 | 0
Blood Potassium Decreased (Investigations) | 1 | 0
Blood Pressure Systolic Increased (Investigations) | 1 | 0
Blood Sodium Decreased (Investigations) | 1 | 0
Blood Uric Acid Increased (Investigations) | 1 | 0
Computerised Tomogram Abdomen Abnormal (Investigations) | 1 | 0
Creatinine Renal Clearance Decreased (Investigations) | 2 | 0
Electrocardiogram Abnormal (Investigations) | 1 | 0
Electrocardiogram Qt Prolonged (Investigations) | 1 | 0
Glycosylated Haemoglobin Increased (Investigations) | 1 | 0
Lipase Increased (Investigations) | 2 | 1
Liver Function Test Abnormal (Investigations) | 1 | 0
Oxygen Saturation Decreased (Investigations) | 1 | 0
Ultrasound Kidney Abnormal (Investigations) | 1 | 0
Waist Circumference Increased (Investigations) | 1 | 0
White Blood Cell Count Decreased (Investigations) | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic Acidosis (Metabolism and nutrition disorders) | 1 | 0
Vitamin D Deficiency (Metabolism and nutrition disorders) | 3 | 1
Aneurysmal Bone Cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 5 | 0
Bone Lesion (Musculoskeletal and connective tissue disorders) | 2 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 2 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral Disc Annular Tear (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint Range Of Motion Decreased (Musculoskeletal and connective tissue disorders) | 3 | 0
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle Mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 5 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteosclerosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 9 | 2
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Soft Tissue Mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendon Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Melanocytic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases To Pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous Cell Carcinoma Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral Cyst (Nervous system disorders) | 1 | 0
Clonus (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Poor Quality Sleep (Nervous system disorders) | 1 | 0
Restless Legs Syndrome (Nervous system disorders) | 3 | 0
Sciatica (Nervous system disorders) | 1 | 0
Sensory Disturbance (Nervous system disorders) | 1 | 0
Viith Nerve Paralysis (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 1
Depression (Psychiatric disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 4 | 1
Panic Attack (Psychiatric disorders) | 1 | 0
Sleep Talking (Psychiatric disorders) | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 2 | 0
Calculus Bladder (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Micturition Urgency (Renal and urinary disorders) | 1 | 0
Nephrocalcinosis (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal Cyst (Renal and urinary disorders) | 1 | 0
Urinary Incontinence (Renal and urinary disorders) | 1 | 0
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0
Testicular Mass (Reproductive system and breast disorders) | 1 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1 | 0
Vulva Cyst (Reproductive system and breast disorders) | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Artery Dilatation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Respiratory Acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Keloid Scar (Skin and subcutaneous tissue disorders) | 1 | 0
Precancerous Skin Lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 0
Rash Papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Irritation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Mass (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Odour Abnormal (Skin and subcutaneous tissue disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 4 | 1
Hypotension (Vascular disorders) | 2 | 0
Peripheral Venous Disease (Vascular disorders) | 1 | 0
Vasodilatation (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2019-09-26): https://cdn.clinicaltrials.gov/large-docs/67/NCT02304367/Prot_000.pdf
  • Statistical Analysis Plan (2016-05-04): https://cdn.clinicaltrials.gov/large-docs/67/NCT02304367/SAP_001.pdf